

# **Study Protocol Cover Page**

Official Study Title: A Phase I/II, Open-label, Dose-escalating, Sequential-cohort Study

Assessing the Safety, Tolerability, Immunogenicity, and Bioactivity of a

Single Intravitreal Injection of DE-122 Injectable Solution for the

Treatment of Refractory Exudative Age-related Macular

Degeneration- PAVE Study

NCT Number: NCT02555306

Date of the document: 30 June 2016

## **DE-122**

## **Protocol 36-001**

### Amendment 03

TITLE: A Phase I/II, Open-label, Dose-escalating, Sequential-cohort Study Assessing the Safety, Tolerability, Immunogenicity, and Bioactivity of a Single Intravitreal Injection of DE-122 Injectable Solution for the Treatment of Refractory Exudative Age-related Macular Degeneration- PAVE Study

| SPONSOR: | STUDY DRUG: |
|---|---|
| SANTEN INCORPORATED<br>2100 Powell Street,<br>16th Floor,<br>Emeryville, CA 94608 | 0.5 mg ( $20\mu L$ of 25 mg/mL) DE-122 injectable solution 1.0 mg ( $40\mu L$ of 25 mg/mL) DE-122 injectable solution 2.0 mg ( $20\mu L$ of 100 mg/mL) DE-122 injectable solution 4.0 mg ( $40\mu L$ of 100 mg/mL) DE-122 injectable solution |

I have read the 36-001 protocol and agree to conduct the study as outlined and in accordance with 21CFR Parts 11, 50, 54, 56, and 312, 42 USC 282 (j), the ethical principles in the Declaration of Helsinki, ICH GCPs, and applicable local regulations. I will not initiate the study until I have obtained written approval by the appropriate Institutional Review Board (IRB) or Ethics Committee (EC) and have complied with all financial and administrative requirements of the governing body of the clinical institution and Santen as the Sponsor. I will obtain written informed consent from each study subject prior to performing any study-specific procedures.

I understand that my electronic signature on an electronic case report form indicates that the data therein has been reviewed and accepted by me as the Investigator. I agree to maintain the confidentiality of all information received or developed in connection with this protocol.

| INVESTIGATOR: | Signature/Date: | | / |
|---------------|-----------------|--------------------|---|
| | Name: | · | |
| | | (Typed or Printed) | |
| | Address: | | |
| | Phone: | | |

# **APPROVERS**



# 1. PROCEDURES IN CASE OF EMERGENCY

**Table 1:** Emergency Contact Information



#### 2. SYNOPSIS

Name of Sponsor/Company: Santen Incorporated

2100 Powell Street, 16<sup>th</sup> Floor Emeryville, CA 94608

Name of Investigational Product: DE-122 injectable solution

Name of Active Ingredient: DE-122, a chimeric anti-CD105 (Endoglin) IgG1 antibody consisting of human  $C\kappa$  and  $C\gamma$ 1 constant regions with murine  $V\kappa$  and  $V_H$  regions

**Title of Study:** A Phase I/II, Open-label, Dose-escalating, Sequential-cohort Study Assessing the Safety, Tolerability, Immunogenicity, and Bioactivity of a Single Intravitreal Injection of DE-122 Injectable Solution for the Treatment of Refractory Exudative Age-related Macular Degeneration - PAVE Study

Estimated date first subject enrolled: August, 2015 Phase I/II

Estimated date last subject completed: April, 2017

#### **Primary Objective:**

• To assess the safety and tolerability of a single intravitreal injection of four dose levels of DE-122 (0.5 mg/eye, 1.0 mg/eye, 2.0 mg/eye and 4.0 mg/eye) in subjects with refractory exudative agerelated macular degeneration.

#### **Secondary Objective:**

• To evaluate the bioactivity of four dose levels of DE-122 in subjects with refractory exudative agerelated macular degeneration.

### Methodology:

This is an open-label, dose-escalating, sequential-cohort study assessing the safety, tolerability, immunogenicity, and bioactivity of a single intravitreal injection of 0.5 mg, 1.0 mg, 2.0 mg and 4.0 mg DE-122 administered in approximately 12 subjects with refractory exudative age-related macular degeneration (AMD).

The subjects will receive a single intravitreal injection of DE-122 in the study eye. The number of subjects will be approximately 12 subjects (2 or 3 subjects in Cohort 1, 3 subjects each in Cohorts 2, 3 and 4). Decisions regarding dose escalation in the next cohort will be based on the recommendations of the Safety Review Team consisting of an external Retina Specialist, the Medical Monitor, and the Drug Safety Physician. Dose-Limiting Toxicity response observed in any cohort will result in termination of the dose escalation.

To be eligible, subjects with refractory exudative AMD in the study eye must have lesions  $\leq 12$  disc areas, contain  $\leq 50\%$  hemorrhage and  $\leq 50\%$  fibrosis and  $\leq 50\%$  retinal pigment epithelial atrophy. Subjects must have received recent Intravitreal Injection of anti-VEGF treatment in the study eye > 30 days and < 60 days prior to Visit 1 (Day 1) and must satisfy all other inclusion and exclusion criteria. Subjects must have best corrected visual acuity (BCVA) of 65 to 20 ETDRS letters (20/50 to 20/400)

The first eligible subject in Cohort 1 will receive a single intravitreal injection of 0.5 mg DE-122 in the study eye and will be evaluated through Visit 3 (Day 8±1). The Safety Review Team will review the safety parameters and determine if the safety and tolerability are acceptable.

If acceptable, up to two additional eligible subjects in Cohort 1 will each receive a single intravitreal

Snellen) in the study eve.

injection of 0.5 mg DE-122 in the study eye before starting Cohort 2. After the first 2 or 3 subjects in Cohort 1 have completed Visit 5 (Day 30±2), the Safety Review Team will review the safety parameters of the first 2 or 3 subjects in Cohort 1 and determine if the next dose (1.0 mg) will be administered to Cohort 2.

The same enrollment procedures will be followed for Cohort 2 (1.0 mg of DE-122), Cohort 3 (2.0 mg of DE-122) and Cohort 4 (4.0 mg of DE-122), however, 3 subjects will be enrolled in these cohorts.

Rescue therapy with anti-VEGF medication may be allowed at Visit 3 (Day 8±1) and/or at Visit 7 (Day 60±3) provided the following rescue criteria are met: < 5 letters gained from baseline BCVA or < 50 microns reduction from baseline central subfield thickness (CST) as measured by spectral-domain optical coherence tomography (SD-OCT).

Subjects who do not receive rescue therapy with anti- VEGF medication at Visit 3 (Day 8±1) will receive anti-VEGF treatment at Visit 5 (Day 30±2).

Anti-VEGF treatment at Visit 5 (Day 30±2) and rescue therapy (at Visit 3 and/or Visit 7) should be performed using the same anti-VEGF medication received just prior to enrollment in the study. Safety assessments will be performed on each subject for up to 90 days.

### **Number of Subjects (planned):**

Approximately 12 subjects (2 or 3 subjects in Cohort 1, 3 subjects each in Cohorts 2, 3 and 4) with refractory exudative age related macular degeneration will be enrolled at 5 sites. The final number of subjects enrolled may be adjusted based on the presence of dose limiting toxicities.

#### **Duration of the Study:**

The duration of this clinical study includes up to a 7-day screening phase and 90-day treatment/ follow-up phase. The subject will receive a single drug injection of DE-122 at Visit 1 (Day 1), if rescue criteria is met, will receive treatment of anti-VEGF medication at Visit 3 (Day 8±1), at Visit 5 (Day 30±2) if not given at Visit 3, and at Visit 7 (Day 60±3) with follow-up for each subject through Day 90.

#### Diagnosis and Main Criteria for Inclusion:

#### **Inclusion Criteria:**

At Screening (Day -7 to Day -1) and Visit 1 (Day 1), subjects must meet all of the following inclusion criteria:

- 1. Provide signed written informed consent on the Institutional Review Board (IRB)/Ethics Committee (EC) approved Informed Consent Form (ICF) and provide authorization as appropriate for local privacy regulations.
- 2. Male or female 50 years of age or older on the date of signing the ICF and able and willing to comply with all treatment and follow-up study procedures.
- 3. Diagnosis of subretinal or intraretinal fluid secondary to exudative age-related macular degeneration as assessed by SD-OCT in the study eye with a minimum of 300  $\mu$ m in the central subfield.
- 4. Prior treatment in the study eye with any intravitreal anti-VEGF medication within the past one year prior to Screening visit (at least 3 anti-VEGF treatments within 6 months or 6 anti-VEGF treatments within 12 months).
- 5. Treatment with intravitreal injection of anti-VEGF > 30 days and < 60 days from Visit 1 (Day 1).
- 6. Clinical examination or imaging shows persistent or increasing lesion activity (intraretinal or

- subretinal fluid, exudation, or hemorrhage) despite continuous anti-VEGF therapy.
- 7. Total lesion size of  $\leq$  12 disc areas, contain  $\leq$  50% hemorrhage and  $\leq$  50% fibrosis and  $\leq$  50% retinal pigment epithelial atrophy in the study eye.
- 8. BCVA of 65 to 20 ETDRS letters (20/50 to 20/400) in the study eye.
- 9. Fellow eye must have BCVA equal to or better than the study eye, but not worse than 35 ETDRS letters (20/200)
- 10. Reasonably clear media and some fixation in the study eye to allow for good quality SD-OCT and fundus photography.

#### **Exclusion Criteria:**

A subject with any of the following conditions is not eligible to participate in the study:

#### Ocular:

- 1. BCVA worse than 20/400 in study eye; worse than 20/200 in fellow eye.
- 2. Use of any of the following treatments or anticipated use of any of the following treatments to the study eye:
  - o Intravitreal or periocular corticosteroid, within 90 days prior to Visit 1 (Day 1) and throughout the study;
  - Fluocinolone acetonide intravitreal implant, within 12 months prior to Visit 1 (Day 1) and throughout the study;
  - Visudyne photodynamic therapy, within 90 days prior to Visit 1 (Day 1) and throughout the study;
- 3. Uncontrolled or advanced glaucoma, evidenced by an intraocular pressure (IOP) of > 21 mmHg or cup/disc ratio > 0.8 while on medical therapy, or chronic hypotony (< 6 mmHg) in the study eye.
- 4. Evidence of any other ocular disease other than exudative age related macular degeneration in the study eye that may confound the outcome of the study (e.g., active diabetic retinopathy, posterior uveitis, pseudovitelliform macular degeneration, moderate/severe myopia).
- 5. History of vitrectomy in the study eye.
- 6. Need for ocular surgery in the study eye during the course of the study.
- 7. YAG laser capsulotomy within 30 days prior to Visit 1 (Day 1) in the study eye.
- 8. Intraocular surgery, including lens removal or laser, within 90 days prior to Visit 1 (Day 1) in the study eye.
- 9. Ocular or periocular infection in either eye.
- 10. Pupillary dilation inadequate for quality stereoscopic fundus photography in the study eye.
- 11. Media opacity that would limit clinical visualization, intravenous fluorescein angiography, or SD-OCT evaluation in the study eye.
- 12. History of herpetic infection in the study eye or adnexa.
- 13. Presence of known active toxoplasmosis, inactive toxoplasmosis or toxoplasmosis scar in

either eye.

14. Presence of any form of ocular malignancy including choroidal melanoma in either eye.

#### Non-Ocular:

- 15. Prior treatment with any agent targeting the endoglin pathway (including a fusion protein that binds bone morphogenic protein).
- 16. Prior treatment with DE-122 injectable solution.
- 17. Use of any of the following treatments or anticipated use of any of the following treatments during the study:
  - a. Systemic treatment with anti-VEGF agents (e.g., bevacizumab)
  - b. Agents targeting the endoglin pathway
- 18. Allergy or hypersensitivity to study drug product, fluorescein dye, or other study related procedures/medications.
- 19. Inadequate renal function: serum creatinine > 1.3 mg/dL and BUN > 2 x the upper limit of normal (ULN).
- 20. Inadequate hematologic function: hemoglobin < 10 g/dL; platelet count < 130 x  $10^9$  /L; WBC < 3.8 X  $10^9$  /L or > 10.9 X  $10^9$  /L.
- 21. Inadequate liver function: serum bilirubin > 1.5 mg/dL, GGT, SGOT/ALT, SGPT/AST, and alkaline phosphatase outside 2 x ULN.
- 22. History of bone marrow suppression.
- 23. Active bleeding or pathologic condition that carries a high risk of bleeding (e.g., hereditary hemorrhagic telangiectasia).
- 24. History of hemorrhage, epistaxis, hemoptysis (> ½ teaspoon bright red blood), or treatment with anticoagulants within 90 days prior to Visit 1 (Day 1).
- 25. Myocardial infarction, stroke or history of transient ischemic attacks within 180 days prior to Visit 1 (Day 1).
- 26. Major surgery within 90 days prior to Visit 1 (Day 1). Major surgery is defined as any surgery involving a risk to the life of the subject, including any operation upon an organ within the cranium, chest, abdomen, or pelvic cavity.
- 27. Therapeutic radiation to the head or neck within 90 days prior to Visit 1 (Day 1).
- 28. Participation in other investigational drug or device clinical trials within 30 days prior to Visit 1 (Day 1) or planning to participate in other investigational drug or device clinical trials for the duration of the study. This includes both ocular and non-ocular clinical trials.
- 29. Uncontrolled blood pressure (defined as systolic > 180 mmHg and/or diastolic > 110 while subject is sitting). If a subject's initial reading exceeds these values, a second reading may be taken 30 or more minutes later. If a subject's blood pressure needs to be controlled by antihypertensive medication, the subject can be eligible if medication is taken continuously for at least 30 days prior to Visit 1 (Day 1).
- 30. Atrial fibrillation not controlled by the subject's primary care physician or cardiologist within

30 days prior to Visit 1 (Day 1).

- 31. Clinically significant concurrent illness, laboratory or EKG abnormality.
- 32. History of other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease condition that contraindicates the use of an investigational drug, might affect the interpretation of the results of the study, or renders the subject at high risk for treatment complications.
- 33. Any systemic infection within 30 days prior to Visit 1 (Day 1).
- 34. Females who are pregnant or lactating and females of child-bearing potential who are not using adequate contraceptive precautions (i.e., IUD, oral contraceptives, barrier method, or other contraception deemed adequate by the Clinical Investigator). Men who do not agree to practice an acceptable method of contraception throughout the course of the study.
- 35. Use of marijuana or illegal medication within 30 days prior to Visit 1 (Day 1) and throughout the study.
- 36. Unable to comply with study procedures or follow-up visits.

In addition, the Clinical Investigator or Santen Medical Monitor may declare a subject ineligible for any sound reason.

#### **Study Eye**

The study eye of an eligible subject is defined as the eye with the worse vision. If both eyes have the same vision, the right eye (OD) should be determined as the study eye.

### Investigational product, dosage and mode of administration:

Subjects will receive one of the following four dose levels of the investigational product, DE-122 injectable solution by intravitreal injection:

- 0.5 mg (20µL of 25 mg/mL) DE-122 injectable solution
- 1.0 mg (40µL of 25 mg/mL) DE-122 injectable solution
- 2.0 mg (20µL of 100 mg/mL) DE-122 injectable solution
- 4.0 mg (40µL of 100 mg/mL) DE-122 injectable solution

#### **Route of Administration of Investigational product:**

Single intravitreal injection in the study eye

#### **Criteria for Evaluation:**

**Safety:** The safety assessments will include adverse events (AEs), slit-lamp biomicroscopy, indirect ophthalmoscopy, BCVA, IOP, fundus photography, fluorescein angiography, serum chemistry, hematology, urinalysis, vital signs, physical exam, EKG and pregnancy.

**Bioactivity:** The bioactivity of DE-122 on resolution of fluid will be assessed using the change in CST based on SD-OCT at each visit post DE-122 treatment as compared to baseline (change in response to anti-VEGF treatment given before Visit 1 (Day 1)).

#### **Statistical Methods:**

In addition to data listings, descriptive summaries will be provided for safety and bioactivity parameters by dose level.

| 3. | TABLE OF CONTENTS, LIST OF TABLES, AND LIST OF FIGURES | |
|----------|--------------------------------------------------------|----|
| 1. | PROCEDURES IN CASE OF EMERGENCY | 3 |
| 2. | SYNOPSIS | 4 |
| 3. | TABLE OF CONTENTS, LIST OF TABLES, AND LIST OF FIGURES | 9 |
| 4. | LIST OF ABBREVIATIONS AND DEFINITIONS OF TERMS | 14 |
| 5. | INTRODUCTION | 16 |
| 6. | OBJECTIVES | 18 |
| 7. | INVESTIGATIONAL PLAN | 19 |
| 7.1. | Overall Study Design and Plan | 19 |
| 7.1.1. | Selection of Concentrations in the Study | 21 |
| 7.2. | Number of Subjects | 21 |
| 7.3. | Treatment Assignment | 21 |
| 7.4. | Dose Adjustment Criteria | 22 |
| 7.4.1. | Safety Criteria for Adjusting or Stopping Doses | 22 |
| 7.5. | Criteria for Study Termination | 23 |
| 7.6. | Study Procedures | 23 |
| 7.6.1. | Screening Phase | 25 |
| 7.6.1.1. | Visit 0/Screening (Day -7 to Day -1) | 25 |
| 7.6.2. | Treatment/follow-up phase | 25 |
| 7.6.2.1. | Visit 1 (Day 1) | 25 |
| 7.6.2.2. | Visit 2 (Day 2) | 27 |
| 7.6.2.3. | Visit 3 (Day 8±1) | 27 |
| 7.6.2.4. | Visit 4 (Day 15±2) | 28 |
| 7.6.2.5. | Visit 5 (Day 30±2) | 29 |
| 7.6.2.6. | Visit 6 (Day 45±3) | 30 |
| 7.6.2.7. | Visit 7 (Day 60±3) | 30 |
| 7.6.3. | Study Exit | 31 |
| 7.6.3.1. | Visit 8/Exit (Day 90±3) | 31 |
| 7.6.4. | Unscheduled Visits | 32 |
| 8. | SELECTION AND WITHDRAWAL OF SUBJECTS | 33 |

| 8.1. | Subject Inclusion Criteria | 33 |
|---|---|---|
| 8.2. | Subject Exclusion Criteria | 33 |
| 8.3. | Subject Withdrawal Criteria | 36 |
| 9. | TREATMENT OF SUBJECTS | 37 |
| 9.1. | Description of Study Drug | 37 |
| 9.2. | Concomitant Medications | 37 |
| 9.2.1. | Prohibited Medications or Treatments | 37 |
| 9.2.2. | Rescue Therapy at Visit 3 (Day 8±1) and/or at Visit 7 (Day 60±3) | 37 |
| 9.2.3. | Anti-VEGF treatment at Visit 5 (Day 30±2) | 37 |
| 9.3. | Treatment Compliance | 38 |
| 9.4. | Randomization and Masking | 38 |
| 10. | STUDY DRUG MATERIALS AND MANAGEMENT | 39 |
| 10.1. | Study Drug | 39 |
| 10.1.1. | Investigational Drug | 39 |
| 10.1.2. | Study Drug Complaint Reporting. | 39 |
| 10.1.3. | Other Study Supplies | 39 |
| 10.2. | Study Drug Packaging and Labeling | 39 |
| 10.3. | Study Drug Storage | 39 |
| 10.4. | Study Drug Preparation | 39 |
| 10.5. | Loading the Syringe. | 40 |
| 10.6. | Eye Preparation | 41 |
| 10.7. | Study Drug Administration | 41 |
| 10.8. | Study Drug Accountability | 42 |
| 10.9. | Study Drug Handling and Disposal | 42 |
| 11. | ASSESSMENT OF SAFETY | 43 |
| 11.1. | Adverse Events | 43 |
| 11.1.1. | Definition of Adverse Events | 43 |
| 11.1.1.1. | Assessment of Adverse Events | 43 |
| 11.1.1.2. | Reporting Adverse Events | 44 |
| 11.1.2. | Serious Adverse Events | 45 |
| 11.1.2.1. | Reporting Serious Adverse Events | 46 |
| 11.1.2.2. | Expedited Reporting of Serious Adverse Events | 46 |
| 11.1.3. | Events of Special Interest. | 46 |

| 11.1.4. | Follow-up of Adverse Events | 47 |
|----------|--------------------------------------------------|----|
| 11.1.5. | Manual Back-Up Reporting Procedures | 47 |
| 11.2. | Safety Parameters | 48 |
| 11.2.1. | Physical Examination | 48 |
| 11.2.2. | Electrocardiogram (EKG) | 48 |
| 11.2.3. | Vital Signs | 48 |
| 11.2.4. | Best Corrected Visual Acuity | 48 |
| 11.2.5. | Slit-lamp Biomicroscopy | 48 |
| 11.2.6. | Intraocular Pressure | 48 |
| 11.2.7. | Indirect Ophthalmoscopy | 48 |
| 11.2.8. | Urine Pregnancy Test | 49 |
| 11.2.9. | Serum Pregnancy Test | 49 |
| 11.2.10. | Serum Chemistry, Hematology and Urinalysis | 49 |
| 11.2.11. | Fundus Photography | 49 |
| 11.2.12. | Fluorescein Angiography | 49 |
| 11.2.13. | Adverse Events | 49 |
| 12. | ASSESSMENT OF BIOACTIVITY | 50 |
| 13. | OTHER ASSESSMENTS | 51 |
| 13.1. | Demographics and Baseline Characteristics | 51 |
| 13.2. | Immunogenicity | 51 |
| 13.3. | Biomarker | 51 |
| 13.4. | Other Assessments | 51 |
| 14. | STATISTICAL METHODS | 52 |
| 14.1. | General Considerations | 52 |
| 14.1.1. | Study Endpoints | 52 |
| 14.1.2. | Sample Size | 52 |
| 14.1.3. | Statistical Hypotheses and Level of Significance | 52 |
| 14.1.4. | Randomization | 52 |
| 14.1.5. | Study Eye | 52 |
| 14.2. | Study Populations | 52 |
| 14.3. | Handling of Missing Values. | 53 |
| 14.5. | Demographics and Baseline Characteristics | 53 |
| 14.6. | Bioactivity Analyses | 53 |

| 14.7. | Safety Analysis | 53 |
|---|---|---|
| 14.8. | Other Analysis | 54 |
| 14.8.1. | Immunogenicity Analysis | 54 |
| 14.8.2. | Biomarker Analysis | 54 |
| 15. | DIRECT ACCESS TO SOURCE DATA/DOCUMENTS | 55 |
| 15.1. | Study Monitoring. | 55 |
| 15.2. | Audits and Inspections | 55 |
| 15.3. | Institutional Review Board | 56 |
| 16. | QUALITY CONTROL AND QUALITY ASSURANCE | 57 |
| 16.1. | Quality Control | 57 |
| 16.2. | Quality Assurance | 57 |
| 17. | ETHICS | 58 |
| 17.1. | Ethics Review | 58 |
| 17.2. | Ethical Conduct of the Study | 58 |
| 17.3. | Written Informed Consent | 58 |
| 18. | DATA HANDLING AND RECORDKEEPING | 59 |
| 18.1. | Inspection of Records | 59 |
| 18.2. | Retention of Records | 59 |
| 18.2.1. | Source Documents | 59 |
| 18.2.2. | Data Collection | 60 |
| 19. | PUBLICATION POLICY | 61 |
| 20. | REFERENCES | 62 |
| 21. | APPENDICES | 64 |
| 21.1. | Appendix A - Obligations of Investigators | 64 |
| 21.2. | Appendix B - Elements of Informed Consent | 66 |
| 21.3. | Appendix C - Declaration of Helsinki | 68 |
| 21.4. | Appendix D - Procedures for Examinations | 74 |
| 21.4.1. | Demographics/Eligibility, Medical/Surgical History and Concomitant Medication | 74 |
| 21.4.2. | Physical Examination | 74 |
| 21.4.3. | Vital Signs | 74 |
| 21.4.4. | EKG | 75 |
| 21.4.5. | Best Corrected Visual Acuity | 75 |

| 21.4.6. | Slit-Lamp Biomicroscopy | 75 |
|-----------|-------------------------------------------------|----|
| 21.4.7. | Intraocular Pressure | 77 |
| 21.4.8. | Indirect Ophthalmoscopy | 78 |
| 21.4.9. | Spectral Domain Optical Coherence Tomography | 78 |
| 21.4.10. | Fundus Photography | 78 |
| 21.4.11. | Fluorescein Angiography | 79 |
| 21.4.12. | Urine Pregnancy Test | 79 |
| 21.4.13. | Serum Pregnancy Test | 79 |
| 21.4.14. | Hematology, Chemistry and Urinalysis | 79 |
| 21.4.15. | Procedure for Immunogenicity Serum Sample | 81 |
| 21.4.16. | Procedure for Biomarker Serum Sample | 81 |
| | LIST OF TABLES | |
| T 11 1 | | 2 |
| Table 1: | Emergency Contact Information | |
| Table 2: | Abbreviations and Specialist Terms | |
| Table 3: | Dose Groups and Associated DE-122 Concentration | |
| Table 4: | Schedule of Events | |
| Table 5: | DE-122 Dosing | |
| Table 6: | Protocol Amendment 03 Summary of Changes | 82 |
| | LIST OF FIGURES | |
| Figure 1: | Study Schematic | 20 |
| Figure 2: | 0.3 mL fill in a 2 mL vial | 40 |
| Figure 3: | Alignment of the syringe (20 µL example) | 41 |

# 4. LIST OF ABBREVIATIONS AND DEFINITIONS OF TERMS

The following abbreviations and specialist terms are used in this study protocol.

**Table 2:** Abbreviations and Specialist Terms

| Abbreviation/Term | Definition |
|---|---|
| ADA | anti-drug antibody |
| AE(s) | adverse event(s) |
| ALT | alanine amino transferase |
| AMD | age-related macular degeneration |
| AST | aspartate amino transferase |
| BCVA | best corrected visual acuity |
| BMP | bone morphogenic protein |
| BUN | blood urea nitrogen |
| CD105 | endoglin |
| CNV | choroidal neovascularization |
| CST | central subfield thickness |
| DE-122 | a chimeric anti-CD105 (endoglin) IgG1 antibody consisting of human C $\kappa$ and C $\gamma$ 1 constant regions with murine V $\kappa$ and V $_{\rm H}$ regions |
| dL | deciliter |
| eCRF(s) | electronic case report form(s) |
| EDC | electronic data capture |
| EKG | Electrocardiogram (= ECG) |
| ETDRS | Early Treatment of Diabetic Retinopathy Study |
| ESI(s) | event(s) of special interest |
| FDA | Food and Drug Administration |
| GCP | Good Clinical Practice |
| GGT | gamma-glutamyl transpeptidase |
| ICF | informed consent form |
| ICH | International Conference on Harmonization |
| IEC | independent ethics committee |
| IOP | intraocular pressure |
| IRB | institutional review board |

 Table 2:
 Abbreviations and Specialist Terms (Continued)

| Abbreviation/Term | Definition |
|-------------------|----------------------------------------------|
| ITT | intention-to-treat |
| IUD | intrauterine device |
| IVT | intravitreal |
| MedDRA | Medical Dictionary for Regulatory Activities |
| mg | milligram |
| μL | microliter |
| mL | milliliter |
| mmHg | millimeter of mercury |
| SAE(s) | serious adverse event(s) |
| SAP | statistical analysis plan |
| SD-OCT | spectral domain optical coherence tomography |
| SGOT | serum glutamic oxaloacetic transaminase |
| SGPT | serum glutamic pyruvic transaminase |
| TGF-β | transforming growth factor-β |
| ULN | upper limit of normal |
| VEGF | vascular endothelial growth factor |

#### 5. INTRODUCTION

AMD is the leading cause of irreversible vision loss in developed countries. AMD is characterized by extracellular matrix deposits, known as drusen, accumulating between the retinal pigment epithelium and Bruch's membrane. In exudative or wet AMD unwanted blood vessels grow into the macula which leads to hemorrhage and subretinal fluid. In addition, retinal pigment epithelial detachment, retinal tears, fibrovascular scarring and vitreous hemorrhage may occur. The aberrant growth of leaky vessels is the result of local inflammatory responses leading to disruption of the balance of cytokines that control angiogenesis (Lim et al., 2008)

Angiogenesis is a complex and coordinated process of the growth and sprouting of new blood vessels from pre-existing vasculature. Although several angiogenic factors have been identified, VEGF family proteins, their receptors and intracellular signaling molecules appear to be the key mediators of angiogenesis (Kane et al., 2008).

Exciting advances have been made in understanding the pathogenesis of AMD in recent years. Since 2004, several anti-VEGF medications, such as ranibizumab (Lucentis®), pegaptanib (Macugen®) and aflibercept (Eylea®) have been approved by the FDA for patients with exudative AMD. Although Eylea®, which is the most recently approved anti-VEGF medication for exudative AMD, showed more than 95% of the subjects maintained vision defined as losing < 15 ETDRS letters for 12 months; however, only 30% of subjects gained > 15 ETDRS letters. Moreover, approximately 30% of subjects still showed cystic intraretinal edema and subretinal fluid after 12 months of treatment (Heier et al., 2012). Therefore, anti-VEGF treatment may not represent the only pathway towards anti-angiogenesis. New or novel approaches to inhibit angiogenesis are needed to elicit further improvements in visual acuity, macular edema, and quality of life in exudative AMD patients.

Endoglin (also known as CD105) is a member of the TGF- $\beta$  receptor family that is expressed by proliferating endothelial cells and is considered as one of the essential factors for angiogenesis. Normal levels of endoglin are needed for endothelial cell proliferation (Guo et al., 2004; Warrington et al., 2005). Endoglin expression is increased by cellular hypoxia through the production of hypoxia-inducible factor-1- $\alpha$  (HIF-1- $\alpha$ ), and endoglin protects hypoxic cells from apoptosis (Li et al., 2003).

Endoglin acts to modulate signaling of multiple kinase receptor complexes of the TGF-β superfamily, including TGF-β receptors, bone morphogenic protein (BMP) receptors, activin receptor-like kinases (ALKs) and activin receptors (Barbara et al., 1999). In the absence of endoglin, activation of TGF-β receptors results in phosphorylation of SMAD 2/3 proteins that inhibit endothelial cell growth. However, activation of endoglin by BMP modulates SMAD protein phosphorylation, through phosphorylation of SMAD 1/5/8 (Nolan-Stevaux et al., 2012). The end result is release of the growth inhibitory effects of TGF-β receptor activation on endothelial cells (Lebrin et al., 2004). Similarly, endoglin is required for proliferation of endothelium in response to BMP. BMP-9 and BMP-10 bind to endoglin to induce phosphorylate SMAD 1/5/8 to signal endothelial cell proliferation (Park et al., 2008).

A recent study has demonstrated that endoglin is highly expressed in choroidal neovascularization (CNV) membranes surgically excised from exudative AMD patients (Yasukawa et al., 2000).

TRC105 is an anti-angiogenic mouse/human chimeric antibody against human endoglin developed by TRACON Pharmaceuticals, Inc. TRC105 binds endoglin on proliferating endothelial cells to inhibit ligand binding by BMP, interrupting signal transduction, resulting in growth inhibition and apoptosis. TRC105 also mediates antibody-dependent cell-mediated cytotoxicity (ADCC).

A series of pharmacology studies in the TRACON oncology program have characterized TRC105 as a potent anti-angiogenic agent. TRC105 alone inhibits VEGF- and bFGF-induced endothelial cell proliferation, suggesting that TRC105 can achieve similar therapeutic effects as anti-VEGF agents but through a different mechanism and specific or shared signaling pathway.

It may be that TRC105 and anti-VEGF agents work synergistically to inhibit neovascularization and TRC105 suppresses the escape mechanism underlying resistance to the long-term anti-VEGF treatment, both of which are mediated by overexpression of endoglin.

Several clinical trials for various cancer patients have being conducted by TRACON Pharmaceuticals, Inc. As of 06 December 2014, over 300 patients had been treated with TRC105. The majority of the patients have been Caucasian with ages ranging from 18-87 years. TRC105 has been well tolerated and exhibited a remarkably consistent adverse event profile, whether dosed as a single agent or dosed in combination with VEGF inhibitors or chemotherapy. Activity of TRC105 in combination has been particularly noteworthy and represents the current development strategy.

Santen is developing an ophthalmic formulation of TRC105 - DE-122 injectable solution - suitable for intravitreal injection for the treatment of exudative AMD.

Santen is opening the IND with this Phase I/II study (Protocol 36-001), open-label, dose-escalating, sequential cohort study assessing the safety, tolerability, immunogenicity, and bioactivity of a single IVT injection of DE-122 injectable solution in the study eye of approximately twelve subjects with refractory exudative AMD. Four dose levels of DE-122 will be assessed in the Phase I/II study; 0.5 mg/eye, 1.0 mg/eye, 2.0 mg/eye and 4.0 mg/eye. The doses selected for use in this study were based on results from the nonclinical studies. Additional information regarding the nonclinical studies is provided in the Investigator's Brochure.

As of June 2016, 2 subjects in Cohort 1 have been enrolled and completed the study with no adverse events, and no safety and tolerability concerns.

## 6. **OBJECTIVES**

## Primary Objective:

• To assess the safety and tolerability of a single intravitreal injection of four dose levels of DE-122 (0.5 mg/eye, 1.0 mg/eye, 2.0 mg/eye and 4.0 mg/eye) in subjects with refractory exudative age-related macular degeneration.

## Secondary Objective:

• To evaluate the bioactivity of four dose levels of DE-122 in subjects with refractory exudative age-related macular degeneration.

#### 7. INVESTIGATIONAL PLAN

## 7.1. Overall Study Design and Plan

This is an open-label, dose-escalating, sequential-cohort study assessing the safety, tolerability, immunogenicity, and bioactivity of a single IVT injection of 0.5 mg, 1.0 mg, 2.0 mg and 4.0 mg DE-122 injection administered in a total of approximately 12 subjects with refractory exudative AMD.

Approximately 12 subjects in four cohorts (2 or 3 subjects in Cohort 1, 3 subjects each in Cohorts 2, 3 and 4) will receive a single IVT injection of DE-122 in the study eye. Decisions regarding dose escalation will be based on the recommendations of the Safety Review Team consisting of an external Retina Specialist, the Medical Monitor, and the Drug Safety Physician. Dose-Limiting Toxicity response observed in any cohort will result in termination of the dose escalation.

The study is designed to include up to a 7-day screening phase and 90-day treatment/follow-up phase for each subject.

The first eligible subject in Cohort 1 will receive a single intravitreal injection of 0.5 mg DE-122 in the study eye and will be evaluated through Visit 3 (Day 8±1). The Safety Review Team will review the safety parameters and determine if the safety and tolerability are acceptable.

If acceptable, up to two additional eligible subjects in Cohort 1 will each receive a single intravitreal injection of 0.5 mg DE-122 in the study eye before starting Cohort 2. After the first 2 or 3 subjects in Cohort 1 have completed Visit 5 (Day 30±2), the Safety Review Team will review the safety parameters of the first 2 subjects in Cohort 1 and determine if the next dose (1.0 mg) will be administered to Cohort 2.

The same enrollment procedures will be followed for Cohort 2 (1.0 mg of DE-122), Cohort 3 (2.0 mg of DE-122) and Cohort 4 (4.0 mg of DE-122), however 3 subjects must be enrolled in these cohorts.

Rescue therapy with anti-VEGF medication may be allowed at Visit 3 (Day 8±1) and/or at Visit 7 (Day 60±3) provided the following rescue criteria are met: < 5 letters gained from baseline BCVA or < 50 microns reduction from baseline CST as measured by SD-OCT.

All subjects will receive IVT anti-VEGF treatment at Visit 5 (Day 30±2) after DE-122 IVT injection, in order to avoid a prolonged period without treatment, if no rescue therapy was given at Visit 3 (Day 8±1), regardless of the visual acuity and CST outcomes.

All anti-VEGF treatment should be performed using the same anti-VEGF medication received just prior to enrollment in the study.

Safety assessments will be performed on each subject for up to 90 days.

All subjects will be closely monitored at Days 8 and/or 30 for dose limiting toxicities by the Safety Review team (Section 7.4.1).

Randomization is not employed in this study due to the small sample size and the dose-escalating design. Refer to Figure 1 for a pictorial representation of the study design.

Figure 1: Study Schematic



### 7.1.1. Selection of Concentrations in the Study

In this clinical study, four dose levels of DE-122 (0.5 mg, 1.0 mg, 2.0 mg or 4.0 mg) are being tested in subjects with refractory exudative AMD. Systemic exposure of DE-122 in this study given by a single IVT injection at dose levels up to 4.0 mg/eye is anticipated to be significantly lower than the systemic exposure in over 300 cancer subjects (most of whom received 10 mg/kg of TRC105 by weekly intravenous infusion). Therefore, no concerns regarding systemic toxicity are anticipated in this study.

In pre-clinical studies, the highest tested DE-122 IVT dose of 5 mg/monkey eye would correlate to 10 mg/eye in human eyes due to the difference in volume, hence the difference in vitreous volume between human and monkey (2:1 ratio) conveys a margin of safety.

The starting IVT dose of 0.5 mg utilized in this clinical study is only 1/10 (10%) of the 5 mg dose determined as safe in the single dose toxicity study in cynomolgus monkeys by IVT injection (and 1/20, or 5%, of the safe 5 mg dose taking into account differences in monkey and human vitreous volumes). The highest 4.0 mg dose tested in this clinical study is only 80% of the safe dose in monkeys (and 40% of that dose with differences in vitreous volume considered).

In the mouse model of laser-induced CNV efficacy study, animals were given an IVT injection of DE-122 at 0.5, 1.5 and 5.0  $\mu$ g/eye. DE-122 inhibited CNV in a dose-dependent manner. The lowest effective dose was 0.5  $\mu$ g/eye. Considering the vitreous volume difference between human and mouse (~1000:1 ratio), 0.5 mg/eye is considered a logical starting dose level for this initial clinical study. In addition, the 0.5 mg DE-122 IVT dose is 10 times lower than the tolerated dose of 5.0 mg/eye utilized in the single dose toxicity study in cynomolgus monkeys, aside from the margin of safety conferred by the difference in vitreous volume between monkey and human eyes described above.

# 7.2. Number of Subjects

Approximately 12 subjects (2 or 3 subjects in Cohort 1, 3 subjects each in Cohorts 2, 3 and 4) with refractory exudative age related macular degeneration will be enrolled at 5 sites. The final number of subjects enrolled may be adjusted based on the presence of dose limiting toxicities.

# 7.3. Treatment Assignment

Four dose levels of DE-122 will be administered by a single IVT injection in the study eye as noted in Table 3.

Table 3: Dose Groups and Associated DE-122 Concentration

| Dose Group | DE-122 Concentration |
|-----------------|------------------------------------|
| Cohort 1: 0.5mg | 20 microliters of 25 mg/mL DE-122 |
| Cohort 2: 1.0mg | 40 microliters of 25 mg/mL DE-122 |
| Cohort 3: 2.0mg | 20 microliters of 100 mg/mL DE-122 |
| Cohort 4: 4.0mg | 40 microliters of 100 mg/mL DE-122 |

## 7.4. Dose Adjustment Criteria

The Safety Review Team will review safety parameters after the first subject in a given cohort has completed Visit 3 (Day 8±1). The remaining subjects in the cohort will receive the same dose if neither the safety criteria for adjusting or stopping doses (Section 7.4.1) nor the criteria for study termination (Section 7.5) preclude their treatment.

When the first 2 or 3 subjects in Cohort 1 and 3 subjects in other Cohorts have completed Visit 5 (Day 30±2), the Safety Review Team will again evaluate the safety parameters. If the safety criteria for adjusting or stopping doses and the criteria for study termination are not met, the first subject in the next cohort will receive the next higher DE-122 dose level.

The same safety evaluations will be performed for each cohort.

## 7.4.1. Safety Criteria for Adjusting or Stopping Doses

If more than one of the following dose limiting toxicities is observed in any one cohort, planned doses may be adjusted or stopped by the Safety Review Team.

- Visual acuity loss from baseline defined as:
  - Loss of best corrected visual acuity (BCVA) of 30 or more letters not due to vitreous hemorrhage or injection procedure **OR**
  - o Transition to no light perception (NLP) not due to injection procedure
- Clinically significant inflammation defined as:
  - > 3+ vitreous haze as measured by the National Eye Institute Grading Scheme (Nussenblatt et al., 1985) OR
  - Sterile endophthalmitis (including the presence of hypopyon)
- Severe IOP elevation as measured by tonometry, on two separate exams, at least one day apart, excluding day of injection (despite pharmaceutical intervention):
  - $\circ$  > 35 mmHg **OR**
  - o Increase of > 15 mmHg from baseline

If any of the following adverse events (AEs) occur in any one subject in any cohort, planned doses will be adjusted by treating additional subjects at the same or lower dose level (the occurrence of a second adverse event in either the same or different subjects in one cohort will qualify for study termination, Section 7.5):

- Retinal non-perfusion of the study eye/vascular occlusion
- Vasculitis
- Retinitis
- > 2+ disc edema
- > 2 quadrants of retinal hemorrhage

If there is insufficient safety information in a given cohort at any time, the Safety Review Team may determine to treat additional subjects within that cohort before moving to the next cohort.

## 7.5. Criteria for Study Termination

Unacceptable safety signals that prevent moving to the next higher dose cohort or result in stopping the study may include any of the following, if deemed to be related to study drug DE-122 (not DE-122 administration procedures):

- Pattern of systemic AEs
- Any of the following AEs in any 2 subjects in any cohort:
  - o Retinal Non-perfusion of the study eye/vascular occlusion
  - Vasculitis
  - o Retinitis
  - $\circ$  > 2+ disc edema
  - > 2 quadrants of retinal hemorrhage

# 7.6. Study Procedures

All subjects must sign a written ICF before participating in any study-related activity. Enrollment will occur at Visit 1 (Day 1) after a subject meets all eligibility requirements at Screening (Day -7 to Day -1) and Visit 1 (Day 1). Each enrolled subject will be assigned a unique subject number. If a subject is discontinued from the study for any reason, the subject number will remain in effect and will not be reused.

A Schedule of Events can be found below and detailed procedures for examinations can be found in Section 21.4, Appendix D – Procedures for Examinations.

**Table 4:** Schedule of Events

| Visit Number | Visit 0<br>(SCRN) | Vi | sit 1 | Visit 2 | Visit 3 | Visit<br>4 | Visit<br>5 | Visit<br>6 | Visit<br>7 | Visit<br>8<br>/Exit |
|---|---|---|---|---|---|---|---|---|---|---|
| Visit Schedule | D-7 | ] | D1 | D2 | D8 | D15 | D30 | D45 | D60 | D90 |
| (Time window; days) | to -1 | Pre | Post | D2 | (±1) | (±2) | (±2) | (±3) | (±3) | (±3) |
| Informed consent <sup>a</sup> | X | | | | | | | | | |
| Demographics/Eligibility | X | X | | | | | | | | |
| Medical/surgical history,<br>Concomitant medication | X | X | | X | X | X | X | X | X | X |
| Physical exam | X | | | | | | | | | X |
| Vital signs | X | X | | X | X | X | X | X | X | X |
| EKG | X | | | | X | | X | | | X |
| BCVA (ETDRS) | X | X | | X | X | X | X | X | X | X |
| Slit-lamp biomicroscopy <sup>b</sup> | X | X | X | X | X | X | X | X | X | X |
| Intraocular pressure <sup>c</sup> | X | X | X | X | X | X | X | X | X | X |
| Indirect ophthalmoscopy <sup>b</sup> | X | X | X | X | X | X | X | X | X | X |
| SD-OCT | X | X | | X | X | X | X | X | X | X |
| Fundus photography | X | | | | | | X | | X | X |
| Fluorescein angiography | X | | | | | | X | | X | X |
| Urine pregnancy test <sup>d</sup> | | | | | | | X | | X | |
| Urinalysis <sup>e</sup> | X | | | | X | | X | | | X |
| Serum pregnancy test <sup>d</sup> | X | | | | | | | | | X |
| Hematology, chemistry serum sample <sup>e</sup> | X | | | | X | | X | | | X |
| Immunogenicity serum sample | | X | | | | | X | | | |
| Biomarker serum sample <sup>f</sup> | | X | | X | X | | X | | | X |
| DE-122 IVT Injection | | | X | | | | | | | |
| Rescue with anti-VEGF Injection <sup>g</sup> | | | | | (X) | | | | (X) | |
| Anti-VEGF Injection <sup>h</sup> | | | | | | | X | | | |
| Adverse events | | X | X | X | X | X | X | X | X | X |

a. Informed Consent Form - obtain prior to conducting any study-related activities.

b. Slit-lamp biomicroscopy and indirect ophthalmoscopy will be performed prior to DE-122 or anti-VEGF intravitreal injection and within 30 minutes after injection.

c. IOP will be performed before DE-122 or anti-VEGF Intravitreal injection and 40±10 minutes after injection. If IOP is increased ≥ 10 mmHg, repeat IOP measurement 60±10 minutes after the injection.

d. Serum and urine pregnancy tests are to be performed on all women of child-bearing potential.

e. Collect fasting urine and blood specimen.

f. Biomarker serum sample will be collected from the subjects in Cohorts 3 and 4.

g. If subjects meet the following rescue criteria at Visit 3 (Day 8±1) and/or at Visit 7 (Day 60±3): <5 letters gained from baseline BCVA or < 50 microns reduction from baseline CST as measured by SD-OCT.

h. Subjects who do not receive rescue therapy with anti-VEGF medication at Visit 3 (Day 8±1) will receive anti-VEGF treatment at Visit 5 (Day 30±2).

### 7.6.1. Screening Phase

## 7.6.1.1. Visit 0/Screening (Day -7 to Day -1)

- Explain the purpose and details of the study to the subject and obtain written informed consent prior to the subject's participation in any study related activity.
- Obtain subject's demographic information, medical, surgical and medication history.
- Perform the following assessments: (all ophthalmic procedures to be performed OU)
  - Physical examination (if not performed by external internist)
  - Vital signs
  - EKG
  - BCVA (ETDRS)
  - Slit-lamp biomicroscopy
  - IOP
  - Indirect ophthalmoscopy
  - SD-OCT
  - Fundus photography
  - Fluorescein angiography
- Review the inclusion and exclusion criteria. <u>Do not</u> continue screening any subject who does not meet the screening eligibility requirements.
- If the subject continues to be eligible for the study, collect more than 8 hours fasting urine and blood specimen for the following examinations:
  - Urinalysis
  - Serum pregnancy test (for females of child-bearing potential)
  - Hematology, chemistry serum sample
- If subject has not been fasting, schedule the subject as soon as possible for fasting blood draw and urine specimen.
- Upload all collected images (SD-OCT, fundus photograph and fluorescein angiogram) to sponsor.
- Schedule the subject to return for Visit 1 (Day 1).

#### 7.6.2. Treatment/follow-up phase

### 7.6.2.1. Visit 1 (Day 1)

• Review results of the following procedures performed at Screening (Day -7 to Day -1) to determine continuation in the study:

- Physical exam
- EKG
- Urinalysis
- Blood chemistry and hematology tests
- Serum pregnancy test (for females of child-bearing potential)
- If the subject continues to be eligible for the study, the following assessments must be performed prior to administration of DE-122 to confirm eligibility and obtain baseline characteristics:
  - Query for AEs
  - Update medical history and medications
  - Vital signs
  - BCVA (ETDRS)
  - Slit-lamp biomicroscopy
  - IOP
  - Indirect ophthalmoscopy
  - SD-OCT
  - Immunogenicity serum sample
  - Biomarker serum sample (in Cohorts 3 and 4)
- Perform final review of inclusion/exclusion criteria. If the subject meets all eligibility criteria, determine the study eye (Section 14.1.5), and then perform DE-122 administration.
- The following procedures must be performed for DE-122 administration (Section 10):
  - Prepare the DE-122 (Section 10.4)
  - Load the syringe (Section 10.5)
  - Prepare the eye including ocular antisepsis of study eye (Section 10.6)
  - Administer DE-122 (Section 10.7)
- The following assessments must be performed after the administration of DE-122:
  - Within 30 minutes following DE-122 injection
    - Slit-lamp biomicroscopy
    - Indirect ophthalmoscopy
  - IOP 40 ( $\pm 10$ ) minutes following DE-122 injection
    - If post-injection IOP is increased  $\geq 10$  mmHg from pre-injection IOP, the IOP will be measured again 60 ( $\pm 10$ ) minutes following injection. If there

is an increase of  $\geq 10$  mmHg at 60 ( $\pm 10$ ) minutes post-injection compared to pre-injection IOP, the subject should be prescribed a topical IOP-lowering medication and monitored for resolution of the event by the Clinical Investigator. An IOP increase of  $\geq 10$  mmHg shall be reported as an AE.

- AE assessments must be performed after the DE-122 administration
- Upload all collected images (SD-OCT) to sponsor.
- Schedule the subject to return for Visit 2 (Day 2).

### 7.6.2.2. Visit 2 (Day 2)

- Perform the following assessments:
  - Query for AEs
  - Update medical history and medications
  - Vital signs
  - BCVA (ETDRS)
  - Slit-lamp biomicroscopy
  - IOP
  - Indirect ophthalmoscopy
  - SD-OCT
  - Biomarker serum sample (in Cohorts 3 and 4)
- Upload all collected images (SD-OCT) to sponsor.
- Instruct the subject to fast for a minimum of 8 hours prior to next visit.
- Schedule the subject to return for the Visit 3 (Day 8±1).

## 7.6.2.3. Visit 3 (Day 8±1)

- Perform the following assessments:
  - Query for AEs
  - Update medical history and medications
  - Vital signs
  - EKG
  - BCVA (ETDRS)
  - Slit-lamp biomicroscopy
  - IOP
  - Indirect ophthalmoscopy

- SD-OCT
- Urinalysis
- Hematology, chemistry serum sample
- Biomarker serum sample (in Cohorts 3 and 4)
- Upload all collected images (SD-OCT) to sponsor.
- Rescue therapy with anti-VEGF medication may be allowed at Visit 3 (Day 8±1) provided the following rescue criteria are met:
  - < 5 letters gained from baseline BCVA OR</p>
  - < 50 microns reduction from baseline CST as measured by SD-OCT.
- Rescue therapy should be performed using the same anti-VEGF medication administered just prior to enrollment in the study. (Section 9.2.2)
- If rescue is performed, the following assessments must be performed after the administration of anti-VEGF treatment:
  - Within 30 minutes following anti-VEGF treatment
    - · Slit-lamp biomicroscopy
    - Indirect ophthalmoscopy
  - IOP:  $40 (\pm 10)$  minutes following injection
    - If post-injection IOP is increased  $\geq 10$  mmHg from pre-injection IOP, the IOP will be measured again 60 ( $\pm 10$ ) minutes following injection. If there is an increase of  $\geq 10$  mmHg at 60 ( $\pm 10$ ) minutes post-injection compared to pre-injection IOP, the subject should be prescribed a topical IOP-lowering medication and monitored for resolution of the event by the Clinical Investigator. An IOP increase of  $\geq 10$  mmHg shall be reported as an AE.
  - AE assessments must be performed after the anti-VEGF medication administration
- Schedule the subject to return for Visit 4 (Day 15±2).

### 7.6.2.4. Visit 4 (Day 15±2)

- Perform the following assessments.
  - Query for AEs
  - Update medical history and medications
  - Vital signs
  - BCVA (ETDRS)
  - Slit-lamp biomicroscopy

- IOP
- Indirect ophthalmoscopy
- SD-OCT
- Instruct the subject to fast for a minimum of 8 hours prior to next visit.
- Schedule the subject to return for Visit 5 (Day 30±2).

### 7.6.2.5. Visit 5 (Day $30\pm 2$ )

- The following assessments must be performed prior to administration of anti-VEGF medication
  - Query for AEs
  - Update medical history and medications
  - Vital signs
  - EKG
  - BCVA (ETDRS)
  - Slit-lamp biomicroscopy
  - IOP
  - Indirect ophthalmoscopy
  - SD-OCT
  - Fundus photography
  - Fluorescein angiography
  - Urinalysis
  - Urine pregnancy test
  - Hematology, chemistry serum sample
  - Immunogenicity serum sample
  - Biomarker serum sample (in Cohorts 3 and 4)
- Upload all collected images (SD-OCT, fundus photograph and fluorescein angiogram) to sponsor.
- Subjects who did not receive rescue therapy with anti-VEGF medication at Visit 3 (Day 8±1) will receive anti-VEGF treatment. The anti-VEGF medication should be performed using the same drug received just prior to enrollment in the study (Section 9.2.3). If the subject received rescue therapy at Visit 3 (Day 8±1), anti-VEGF treatment and post-injection assessments are not necessary.
- The following assessments must be performed after the administration of anti-VEGF treatment:

- Within 30 minutes following anti-VEGF treatment
  - · Slit-lamp biomicroscopy
  - Indirect ophthalmoscopy
- IOP:  $40 (\pm 10)$  minutes following injection
  - · If post-injection IOP is increased  $\geq 10$  mmHg from pre-injection IOP, the IOP will be measured again 60 ( $\pm 10$ ) minutes following injection. If there is an increase of  $\geq 10$  mmHg at 60 ( $\pm 10$ ) minutes post-injection compared to pre-injection IOP, the subject should be prescribed a topical IOP-lowering medication and monitored for resolution of the event by the Clinical Investigator. An IOP increase of  $\geq 10$  mmHg shall be reported as an AE.
- AE assessments must be performed after the anti-VEGF treatment.
- Schedule the subject to return for Visit 6 (Day 45±3).

### 7.6.2.6. Visit 6 (Day $45\pm 3$ )

- Perform the following assessments:
  - Query for AEs
  - Update medical history and medications
  - Vital signs
  - BCVA (ETDRS)
  - Slit-lamp biomicroscopy
  - IOP
  - Indirect ophthalmoscopy
  - SD-OCT
- Upload all collected images (SD-OCT) to sponsor.
- Schedule the subject to return for Visit 7 (Day 60±3).

### 7.6.2.7. Visit 7 (Day $60\pm3$ )

- Perform the following assessments:
  - Query for AEs
  - Update medical history and medications
  - Vital signs
  - BCVA (ETDRS)
  - Slit-lamp biomicroscopy
  - IOP

- Indirect ophthalmoscopy
- SD-OCT
- Fundus photography
- Fluorescein angiography
- Urine pregnancy test
- Upload all collected images (SD-OCT, fundus photograph and fluorescein angiogram) to sponsor.
- Rescue therapy with anti-VEGF medication may be allowed at Visit 7 (Day 60±3) provided the following rescue criteria are met:
  - < 5 letters gained from baseline BCVA OR</p>
  - < 50 microns reduction from baseline CST as measured by SD-OCT.</li>
- Rescue therapy should be performed using the same anti-VEGF medication administered just prior to enrollment in the study (Section 9.2.2).
- If rescue is performed, the following assessments must be performed after the administration of anti-VEGF treatment:
  - Within 30 minutes following anti-VEGF treatment
    - Slit-lamp biomicroscopy
    - · Indirect ophthalmoscopy
  - IOP:  $40 (\pm 10)$  minutes following injection
    - If post-injection IOP is increased ≥ 10 mmHg from pre-injection IOP, the IOP will be measured again 60 (±10) minutes following injection. If there is an increase of ≥ 10 mmHg at 60 (±10) minutes post-injection compared to pre-injection IOP, the subject should be prescribed a topical IOP-lowering medication and monitored for resolution of the event by the Clinical Investigator. An IOP increase of ≥ 10 mmHg shall be reported as an AE.
  - AE assessments must be performed after the anti-VEGF treatment
- Instruct the subject to fast for a minimum of 8 hours prior to next visit.
- Schedule the subject to return for Visit 8/Exit (Day 90±3).

#### **7.6.3. Study Exit**

#### 7.6.3.1. Visit 8/Exit (Day 90±3)

- Perform the following assessments:
  - Query for AEs
  - Update medical history and medications

- Physical exam (if not performed by external internist)
- Vital signs
- EKG
- BCVA (ETDRS)
- Slit-lamp biomicroscopy
- IOP
- Indirect ophthalmoscopy
- SD-OCT
- Fundus photography
- Fluorescein angiography
- Urinalysis
- Serum pregnancy test (for females of child-bearing potential)
- Hematology, chemistry serum sample
- Biomarker serum sample (in Cohorts 3 and 4)
- Upload all collected images (SD-OCT, fundus photograph and fluorescein angiogram) to sponsor.
- Exit subject from study.

### 7.6.4. Unscheduled Visits

If a subject requires evaluation between scheduled visits, complete all applicable study specified procedures as necessary and record the information on the Unscheduled Visit form.

#### 8. SELECTION AND WITHDRAWAL OF SUBJECTS

Eligible subjects must meet all eligibility criteria described in Section 8.1 and Section 8.2.

## 8.1. Subject Inclusion Criteria

At Screening (Day -7 to Day -1) and Visit 1 (Day 1), subjects must meet all of the following inclusion criteria:

- 1. Provide signed written informed consent on the IRB / EC approved ICF and provide authorization as appropriate for local privacy regulations.
- 2. Male or female 50 years of age or older on the date of signing the ICF and able and willing to comply with all treatment and follow-up study procedures.
- 3. Diagnosis of subretinal or intraretinal fluid secondary to exudative AMD as assessed by SD-OCT in the study eye with a minimum of 300 µm in the central subfield.
- 4. Prior treatment in the study eye with any intravitreal anti-VEGF medication within the past one year prior to Screening visit (at least 3 anti-VEGF treatments within 6 months or 6 anti-VEGF treatments within 12 months).
- 5. Treatment with intravitreal injection of anti-VEGF > 30 days and < 60 days from Visit 1 (Day 1).
- 6. Clinical examination or imaging shows persistent or increasing lesion activity (intraretinal or subretinal fluid, exudation, or hemorrhage) despite continuous anti-VEGF therapy.
- 7. Total lesion size of  $\leq$  12 disc areas, contain  $\leq$  50% hemorrhage and  $\leq$  50% fibrosis and  $\leq$  50% retinal pigment epithelial atrophy in the study eye.
- 8. BCVA of 65 to 20 ETDRS letters (20/50 to 20/400) in the study eye.
- 9. Fellow eye must have BCVA equal to or better than the study eye, but not worse than 35 ETDRS letters (20/200)
- 10. Reasonably clear media and some fixation in the study eye to allow for good quality SD-OCT and fundus photography.

# 8.2. Subject Exclusion Criteria

A subject with any of the following conditions is not eligible to participate in the study:

#### Ocular:

- 1. BCVA worse than 20/400 in study eye; worse than 20/200 in fellow eye.
- 2. Use of any of the following treatments or anticipated use of any of the following treatments to the study eye:
  - o Intravitreal or periocular corticosteroid, within 90 days prior to Visit 1 (Day 1) and throughout the study;

- Fluocinolone acetonide intravitreal implant, within 12 months prior to Visit 1 (Day 1) and throughout the study;
- Visudyne photodynamic therapy, within 90 days prior to Visit 1 (Day 1) and throughout the study;
- 3. Uncontrolled or advanced glaucoma, evidenced by an intraocular pressure (IOP) of > 21 mmHg or cup/disc ratio > 0.8 while on medical therapy, or chronic hypotony (< 6 mmHg) in the study eye.
- 4. Evidence of any other ocular disease other than exudative AMD in the study eye that may confound the outcome of the study (e.g., active diabetic retinopathy, posterior uveitis, pseudovitelliform macular degeneration, moderate/severe myopia).
- 5. History of vitrectomy in the study eye.
- 6. Need for ocular surgery in the study eye during the course of the study.
- 7. YAG laser capsulotomy within 30 days prior to Visit 1 (Day 1) in the study eye.
- 8. Intraocular surgery, including lens removal or laser, within 90 days prior to Visit 1 (Day 1) in the study eye.
- 9. Ocular or periocular infection in either eye.
- 10. Pupillary dilation inadequate for quality stereoscopic fundus photography in the study eye.
- 11. Media opacity that would limit clinical visualization, intravenous fluorescein angiography, or SD-OCT evaluation in the study eye.
- 12. History of herpetic infection in the study eye or adnexa.
- 13. Presence of known active toxoplasmosis, inactive toxoplasmosis or toxoplasmosis scar in either eye.
- 14. Presence of any form of ocular malignancy including choroidal melanoma in either eye.

#### Non-Ocular:

- 15. Prior treatment with any agent targeting the endoglin pathway (including a fusion protein that binds bone morphogenic protein).
- 16. Prior treatment with DE-122 injectable solution.
- 17. Use of any of the following treatments or anticipated use of any of the following treatments during the study:
  - a. Systemic treatment with anti-VEGF agents (e.g., bevacizumab)
  - b. Agents targeting the endoglin pathway
- 18. Allergy or hypersensitivity to study drug product, fluorescein dye, or other study related procedures/medications.
- 19. Inadequate renal function: serum creatinine > 1.3 mg/dL and BUN > 2 x the ULN.
- 20. Inadequate hematologic function: hemoglobin < 10 g/dL; platelet count < 130 x  $10^9$  /L; WBC < 3.8 X  $10^9$  /L or > 10.9 X  $10^9$  /L.

- 21. Inadequate liver function: serum bilirubin > 1.5 mg/dL, GGT, SGOT/ALT, SGPT/AST, and alkaline phosphatase outside 2 x ULN.
- 22. History of bone marrow suppression.
- 23. Active bleeding or pathologic condition that carries a high risk of bleeding (e.g., hereditary hemorrhagic telangiectasia).
- 24. History of hemorrhage, epistaxis, hemoptysis (> ½ teaspoon bright red blood), or treatment with anticoagulants within 90 days prior to Visit 1 (Day 1).
- 25. Myocardial infarction, stroke or history of transient ischemic attacks within 180 days prior to Visit 1 (Day 1).
- 26. Major surgery within 90 days prior to Visit 1 (Day 1). Major surgery is defined as any surgery involving a risk to the life of the subject, including any operation upon an organ within the cranium, chest, abdomen, or pelvic cavity.
- 27. Therapeutic radiation to the head or neck within 90 days prior to Visit 1 (Day 1).
- 28. Participation in other investigational drug or device clinical trials within 30 days prior to Visit 1 (Day 1) or planning to participate in other investigational drug or device clinical trials for the duration of the study. This includes both ocular and non-ocular clinical trials.
- 29. Uncontrolled blood pressure (defined as systolic > 180 mmHg and/or diastolic > 110 while subject is sitting). If a subject's initial reading exceeds these values, a second reading may be taken 30 or more minutes later. If a subject's blood pressure needs to be controlled by antihypertensive medication, the subject can be eligible if medication is taken continuously for at least 30 days prior to Visit 1 (Day 1).
- 30. Atrial fibrillation not controlled by the subject's primary care physician or cardiologist within 30 days prior to Visit 1 (Day 1).
- 31. Clinically significant concurrent illness, laboratory or EKG abnormality.
- 32. History of other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease condition that contraindicates the use of an investigational drug, might affect the interpretation of the results of the study, or renders the subject at high risk for treatment complications.
- 33. Any systemic infection within 30 days prior to Visit 1 (Day 1).
- 34. Females who are pregnant or lactating and females of child-bearing potential who are not using adequate contraceptive precautions (i.e., IUD, oral contraceptives, barrier method, or other contraception deemed adequate by the Clinical Investigator). Men who do not agree to practice an acceptable method of contraception throughout the course of the study.
- 35. Use of marijuana or illegal medication within 30 days prior to Visit 1 (Day 1) and throughout the study.
- 36. Unable to comply with study procedures or follow-up visits.
In addition, the Clinical Investigator or Santen Medical Monitor may declare a subject ineligible for any sound reason.

# 8.3. Subject Withdrawal Criteria

An early termination occurs when a subject who provides written informed consent ceases participation in the study, regardless of circumstances, before the completion of the study. Subjects may voluntarily withdraw from the study at any time for any reason. In addition, the Clinical Investigator or the Medical Monitor may terminate a subject's study participation for reasons related to the best interest of the subject. Subjects who terminate from the study may be replaced. Subjects may be terminated from the study due to any of the following reasons:

- Non-compliance
- Lost to follow-up
- Protocol violation
- Withdrawal by subject
- AEs
- Death
- Other

If a subject is discontinued from the study before completing Visit 8/Exit (Day 90±3), then to the extent possible, all assessments, including safety, that are scheduled to be performed at Visit 8/Exit should be performed on the day of discontinuation.

Subjects who discontinue prematurely may be replaced.

#### 9. TREATMENT OF SUBJECTS

# 9.1. Description of Study Drug

DE-122 is a chimeric anti-CD105 IgG1 antibody consisting of human  $C\kappa$  and  $C\gamma1$  constant regions with murine  $V\kappa$  and  $V_H$  regions. DE-122 is composed of two light chains of 213 amino acids and two heavy chains of 448 amino acids and has an approximate molecular weight of 148 kDa. DE-122 is utilized in this clinical study in a formulation designed for IVT injection.

#### 9.2. Concomitant Medications

The use of any concomitant prescription or over-the-counter medication will be recorded during the study. Therapy considered necessary for the subject's welfare may be given at the discretion of the Clinical Investigator during the study. Whenever possible, concomitant medications should be administered in dosages that remain constant throughout the study. The generic name, indication, route of administration, frequency, dose, start date and stop date (if applicable) will be recorded for each medication.

#### 9.2.1. Prohibited Medications or Treatments

Any treatments for exudative AMD in the study eye other than DE-122 are prohibited during the study, except anti-VEGF treatment as a rescue therapy at Visit 3 (Day  $8\pm1$ ) and/or at Visit 7 (Day  $60\pm3$ ), and anti-VEGF treatment at Visit 5 (Day  $30\pm2$ ) as described in Section 9.2.2 and Section 9.2.3.

Any systemic treatments with anti-VEGF agents (e.g., bevacizumab) are prohibited during the study.

The decision to administer a prohibited concomitant medication or treatment during the study should be made with the safety of the subject as the primary consideration. Whenever possible, Santen should be notified before any prohibited medication or treatment is administered or if the permissibility of a specific medication or treatment is in question.

#### 9.2.2. Rescue Therapy at Visit 3 (Day 8±1) and/or at Visit 7 (Day 60±3)

Rescue therapy is defined as IVT injection of anti-VEGF medication which is the same medication administered just prior to the enrollment in the study. Rescue therapy with anti-VEGF medication may be allowed at Visit 3 (Day 8±1) and/or at Visit 7 (Day 60±3) provided the following rescue criteria are met: < 5 letters gained from baseline BCVA or < 50 microns reduction from baseline CST as measured by SD-OCT.

#### 9.2.3. Anti-VEGF treatment at Visit 5 (Day 30±2)

Subjects who did not receive rescue therapy with anti-VEGF medication at Visit 3 (Day 8±1) will receive anti-VEGF treatment at Visit 5 (Day 30±2). The anti-VEGF injection should be performed using the same anti-VEGF medication administered just prior to the enrollment in the study.

# 9.3. Treatment Compliance

In order to obtain reliable safety and bioactivity data, it is critical that the treatment regimen and visit schedule specified in this protocol are followed. The Clinical Investigator is required to administer the DE-122 injection and is responsible for scheduling the subject for follow-up visits as specified in the protocol. Study monitors will verify pertinent data to confirm the study is conducted according to the protocol.

# 9.4. Randomization and Masking

Randomization is not employed in this study due to the small sample size and the open-label, dose-escalating design.

#### 10. STUDY DRUG MATERIALS AND MANAGEMENT

# 10.1. Study Drug

#### 10.1.1. Investigational Drug

DE-122 for IVT injection is formulated in a proprietary, clear, aqueous solution at two concentrations. The 4 dose levels of DE-122 to be administered in the study eye are shown in Table 5.

Table 5: DE-122 Dosing

| Injection Volume of: | Will deliver approximately: |
|------------------------------------|-----------------------------|
| 20 microliters of 25 mg/mL DE-122 | 0.5 mg DE-122 |
| 40 microliters of 25 mg/mL DE-122 | 1.0 mg DE-122 |
| 20 microliters of 100 mg/mL DE-122 | 2.0 mg DE-122 |
| 40 microliters of 100 mg/mL DE-122 | 4.0 mg DE-122 |

The Clinical Investigator will use syringes and needles supplied by Santen/Representative.

#### 10.1.2. Study Drug Complaint Reporting

Complaints regarding the DE-122 for IVT injection should be reported to Santen/Representative Product Complaint at 415-268-9100.

#### 10.1.3. Other Study Supplies

Laboratory supplies for obtaining blood and urine specimens will be supplied by the central laboratory. Santen/Representative will supply a fluoroquinolone equivalent antibiotic eye drop, 10% povidone iodine, needles, and syringes.

# 10.2. Study Drug Packaging and Labeling

DE-122 injectable solutions are filled (0.3 mL fill) in 2-mL Type 1 Glass (borosilicate) clear vials, capped with 13 mm Gray Butyl stoppers with B2-40 coating, and sealed with a 13 mm colored Flip-Off Truedge. Each single use vial will be placed in a unit carton, and the labeling will include protocol number, kit number, and storage conditions.

# 10.3. Study Drug Storage

DE-122 injectable solutions will be provided by Santen/Representative and will be stored in an appropriate secure area at the investigational site. DE-122 vials should be protected from light, stored upright, and kept refrigerated at 2° to 8°C (36° to 46°F).

# 10.4. Study Drug Preparation

<Investigational drug: DE-122>

Once an investigational drug vial number has been assigned to the subject, the vial of investigational drug with the assigned vial number will be removed from the refrigerator. Care should be taken to protect the product from light. Investigational drug should be drawn into the provided sterile single-use custom marked syringe (see Section 10.5) within 30 minutes after removing the vial from the refrigerator. Investigational drug should be injected within 1 hour of being drawn up into the single-use syringe.

Each vial contains enough DE-122 to inject one subject. Each vial will be used one time only.

## 10.5. Loading the Syringe

<Investigational drug: DE-122>

A sterile, single-use 250  $\mu$ L syringe custom marked at 20  $\mu$ L or 40  $\mu$ L will be provided separately for IVT injection of DE-122. Instructions for filling the syringe are as follows:

- 37. Remove the sterile, single-use 250  $\mu$ L syringe, custom marked at 20  $\mu$ L or 40  $\mu$ L, from the packaging.
- 38. Attach a 19-gauge x 1 ½ inch filter needle to the syringe. DE-122 is dispensed in a 0.3 ml fill in a 2mL vial. See Figure 2.
- 39. Using sterile technique, carefully draw up approximately 200  $\mu$ L of DE-122 into the syringe. (Sufficiently larger volume than 20 or 40  $\mu$ L is needed to allow for dead space in syringe and needles prior to IVT injection).
- 40. Remove the 19-gauge x 1½ inch filter needle from the syringe and replace with a 30-gauge x 0.5 inch needle for the IVT injection.
  - a. Ensure that the 30-gauge x 0.5 inch needle is affixed tightly to the syringe.
  - b. Align the top edge of the red O-ring of the plunger with the  $20~\mu L$  or  $40\mu L$  black mark on the syringe, expelling the excess fluid drawn up. See Figure 3.
  - c. Ensure there are no air bubbles within the syringe or the needle hub prior to injection, and prior to expelling the excess fluid drawn up.

Figure 2: 0.3 mL fill in a 2 mL vial





Figure 3: Alignment of the syringe (20 μL example)



# 10.6. Eye Preparation

<Investigational drug: DE-122>

Prior to DE-122 administration, the study eye should be prepared as follows:

- 1. Dilate pupil (1% mydriacyl and 2.5% phenylephrine or equivalent applied topically) approximately 10 minutes prior to injection.
- 2. Administer 1 eye drop of topical anesthetic (0.5% proparacaine hydrochloride ophthalmic solution or an equivalent topical ophthalmic anesthetic).
- 3. Administer 10% povidone iodine.
- 4. Use a sterile cotton-tipped applicator to remove excess fluid from the lower conjunctival sac.
- 5. Take 2 sterile cotton tipped applicators and thoroughly soak with 0.5% proparacaine topical anesthetic eye drops or an equivalent topical ophthalmic anesthetic. Place the soaked applicators, side by side, gently but firmly on the conjunctival surface at the area of the entry site described below in Step 2 (Section 10.7) and hold in place for approximately 1 minute.
- 6. Insert sterile eyelid speculum.
- 7. Place sterile eye drape over study eye.

<Rescue with anti-VEGF medication at Visit 3/Visit 7 or anti-VEGF treatment at Visit 5>

Eye preparation for anti-VEGF administration to be done as per anti-VEGF drug labeling or standard manner in the clinical site.

# **10.7.** Study Drug Administration

<Investigational drug: DE-122>

1. Prior to starting the injection procedure, DE-122 should have been prepared as described in Section 10.4 and Section 10.5, and the study eye should have been prepared as described in Section 10.6.

- 2. If the subject is phakic, the entry site is 4.0 mm from the limbus. If the subject is pseudophakic or aphakic, the entry site is 3.5 mm from the limbus. A caliper may be used to identify the needle entry site.
- 3. Insert the needle perpendicular to the eye wall at the location specified in Step 2 (Section 10.7). The needle should be inserted until the tip is just visible through the dilated pupil. Note: If paracentesis is considered necessary, it should be performed prior to injection of the DE-122 and noted in the source documents.
- 4. Very slowly, inject the entire DE-122 dose volume (20  $\mu$ L or 40  $\mu$ L) and slowly withdraw the needle. Do not pull back on the plunger at any time prior to withdrawing the needle.
- 5. Briefly apply pressure for approximately 1 minute to the needle entry site with sterile cotton tipped applicator (may be skipped per Clinical Investigator's discretion).
- 6. Remove the eyelid speculum.
- 7. Patch the study eye at the Clinical Investigator's discretion.
- 8. Prescribe fluoroquinolone equivalent antibiotic eye drops three times/day for two days following injection, to be initiated as soon as possible.

<Rescue with anti-VEGF medication at Visit 3/Visit 7 or anti-VEGF treatment at Visit 5>

The administration procedure for anti-VEGF medication should follow the anti-VEGF drug labeling or standard practice at the clinical site.

# 10.8. Study Drug Accountability

The Principal Investigator is responsible for ensuring that an inventory is conducted upon receipt of the clinical supplies. The temperature recorder from the shipment will be deactivated and authorized study staff will verify that the temperature was maintained at 2° to 8°C (36° to 46°F) during transit. The clinical supplies shipment form should be completed, signed, and returned as directed. A copy must be maintained at the site for the Principal Investigator's records. The Principal Investigator will keep a current record of the inventory, storage conditions and dispensing of all study drugs. This record will be made available to Santen (or designee) for the purpose of accounting for all clinical supplies. Any significant discrepancy and/or deficiency must be recorded with an explanation.

All supplies sent to the Principal Investigator must be accounted for and in no case will study drugs be used in any unauthorized situation. It is the responsibility of the Principal Investigator to ensure that any used and unused supplies are available to Santen (or designee) throughout the study.

# 10.9. Study Drug Handling and Disposal

All investigational products including unused vials of DE-122 supplied by Santen/Representative will be fully accounted for by the monitor with the help of the person responsible for dispensing the DE-122 and will be returned to Santen/Representative or designee. Accountability will be documented by use of drug accountability forms.

The used vials of DE-122 will be stored at the investigational site upon completion of accountability procedures and returned to Santen or designee after the trial is completed.

#### 11. ASSESSMENT OF SAFETY

#### 11.1. Adverse Events

#### 11.1.1. Definition of Adverse Events

An AE is any untoward medical occurrence in a subject administered a pharmaceutical product and which does not necessarily have a causal relationship with DE-122. An AE, therefore, can be an unintended sign (including an abnormal laboratory finding), symptom, or disease that has clinical significance and is temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.

In clinical studies, an undesirable medical condition occurring at any time, including baseline or pre-treatment period, may be recorded as an AE even if no DE-122 has been administered.

Any significant adverse change in a subject's condition from baseline, regardless of causality, is to be considered an AE, unless the change is determined to be a continuation of a pre-existing condition that is documented in the subject's medical history. However, a clinically significant worsening in severity, intensity, or frequency of a pre-existing condition may indicate an AE. In addition, all conditions that lead to hospitalizations, defined as an overnight hospital stay, are considered as AEs. This includes planned elective surgeries.

Lack of efficacy of the IVT DE-122 for the condition being investigated is not considered an AE unless a clinically significant change is assessed by the Clinical Investigator. An elective surgical procedure scheduled or planned prior to study entry is not considered an AE if an overnight hospital stay is not required, and the underlying diagnosis for which surgery is to be performed should be captured in the medical history as a pre-existing condition. The surgical procedure should also include the term "elective" in all reports.

#### 11.1.1.1. Assessment of Adverse Events

Clinical Investigators will seek information on AEs at each subject contact. Subjects should be asked, using a general, non-direct question, if there has been any change in their general health. Direct questioning and examination should then be performed as appropriate.

Severity of the AE should be assessed according to the following criteria:

**Mild:** No interference with the subject's daily activities; no medical intervention/therapy required

**Moderate:** Possible interference with the subject's daily activities; no or minimal medical intervention/therapy required

**Severe:** Considerable interference with the subject's daily activities; medical intervention/therapy required

Regardless of severity, some AEs may also meet regulatory serious criteria. Refer to definitions and reporting of serious adverse events (SAEs) in Section 11.1.2.

A Clinical Investigator who is qualified in medicine must make the determination of the relationship of the investigational drug, DE-122 to each AE (related or not related). The Clinical

Investigator should decide whether, in his or her medical judgment, there is a reasonable possibility that the DE-122 caused the AE/SAE based on facts, evidence, scientific rationales, and clinical judgment. When assessing causality, the Clinical Investigator may consider the following information when determining the relationship to the DE-122 for each AE: mechanism of action, biologic plausibility, confounding risk factors (i.e., medical history, concomitant medications), temporal relationship, dechallenge/rechallenge, and lack of alternative explanation. It should be specified if the AE is related to the injection procedure and not the study drug.

- The AE may be recorded as **Related** to DE-122 if there is a plausible temporal relationship between the onset of the AE and administration of the DE-122, and the AE cannot be readily explained by the subject's clinical state, concurrent illness, or concomitant therapies; and/or the AE follows a known pattern of response to the DE-122; and/or the AE abates or resolves upon discontinuation of the DE-122.
- Reporting the AE as **Not Related** to DE-122 may be considered if, for example, there is good evidence that the AE has an etiology other than the DE-122 (e.g., pre-existing medical condition, underlying disease, concurrent illness, or concomitant medication); and/or the AE has no plausible temporal relationship to administration of the DE-122 (e.g., cancer diagnosed 2 days after dose of DE-122).

## 11.1.1.2. Reporting Adverse Events

AEs, whether spontaneously reported by the subject or noted by authorized study personnel, will be recorded in the subject's medical record and on the appropriate AE eCRF. Each recorded AE will be described by its duration (i.e., start and end dates), severity, regulatory seriousness criteria if applicable, suspected relationship to the DE-122, actions taken and outcome.

AEs that occur after any subject has provided written informed consent, before treatment, during treatment, or within 30 days following the cessation of treatment, whether or not they are related to the study, must be recorded. To improve the quality and precision of acquired AE data, Clinical Investigators should observe the following guidelines:

- Whenever possible, use recognized medical terms when recording. Do not use colloquialisms and/or abbreviations.
- If known, record the diagnosis (i.e., disease or syndrome) rather than component signs and symptoms and /or laboratory or test findings (e.g., record congestive heart failure rather than dyspnea, rales, and cyanosis, and enlarged heart on chest x-ray). However, other events that are considered unrelated to an encountered syndrome or disease should be recorded as individual AEs (e.g., if congestive heart failure and severe headache are observed at the same time and are clinically unrelated, each event should be recorded as an individual AE).
- If the diagnosis is not known, then record the leading component sign, symptom or test finding and describe the other clinically related findings in the narrative description of the case. A suspected diagnosis can be used and described as such (e.g., record suspected or probable myocardial infarction); this has to be updated in the clinical database once the diagnosis is confirmed.

AEs occurring secondary to other events (e.g., sequelae) should be identified by the primary cause. A primary AE, if clearly identifiable, generally represents the most accurate clinical term. If a primary AE is recorded, events occurring secondary to the primary event should be described in the narrative description of the case. For example:

The subject developed orthostatic hypotension and subsequently fainted and fell to the floor wherein she experienced a head trauma and neck pain.

The primary AE in this example is orthostatic hypotension. The fall, head trauma and neck pain should be described in the narrative description of the case.

- For intermittent events (e.g., intermittent headache), the event onset date should be recorded as the date the subject first started to experience the event and resolution date should reflect when the last occurrence resolved or stopped. Separate AEs for each event should not be recorded. For example, if a subject experienced headache on 14SEP2015 lasting for three hours, then subsequently experienced intermittent episodes of headache every day for approximately 3 hours until 21SEP2015, then the AE date of onset is 14SEP2015 and the resolution date is 21SEP2015.
- For intermittent events, record the maximum severity of the individual events. For example, if a subject complains of intermittent headaches for one week and the severity of each headache ranges from mild to moderate, then the severity would be moderate
- For intermittent hospitalizations occurring for a primary AE (e.g., in a subject with multiple sclerosis, commonly known for its relapsing and remitting course, in some cases leading to multiple hospital confinements), the subsequent hospitalizations should be described in the narrative description of the case.
- If treatment was initiated, include the treatment and duration of the medication(s) in the eCRF.

#### 11.1.2. Serious Adverse Events

SAEs are defined as any findings that suggest a significant hazard, contraindication, side effect, or precaution. Any adverse event is considered a serious adverse event if it results in any of the following outcomes:

- Death
- Life threatening:

A life-threatening event is any event that places the subject at immediate risk of death from the event as it occurred; it does not refer to an event that hypothetically might have caused death if it were more severe.

- Hospitalization, at the minimum an overnight stay
- A persistent or significant disability/incapacity
- A congenital anomaly/birth defect

• Other medically significant events:

Other medically significant events are events that may not result in death, be life-threatening, or require hospitalization but may be considered a serious adverse drug experience when, based upon appropriate medical judgment, they may jeopardize the subject and may require medical or surgical intervention to prevent one of the outcomes listed above.

• Sight threatening event:

A sight-threatening event is any event that places the subject at immediate risk of permanently losing vision in either eve as a direct result of the event.

## 11.1.2.1. Reporting Serious Adverse Events

A SAE eCRF must be completed with as much information available within 24 hours of knowledge of the event.

To improve the quality and precision of acquired SAE data, Clinical Investigators should observe the following guidelines:

- **Death** Death is an outcome of an event. The event that resulted in the death should be recorded and reported as a SAE.
- Hospitalizations for Surgical or Diagnostic Procedures The illness leading to the surgical or diagnostic procedure should be recorded as the SAE, not the procedure itself. The procedure should be captured in the case narrative as part of the action taken in response to the illness.

When new significant information (including the outcome of the event) is obtained, the Clinical Investigator should enter the information directly into the eCRF within 24 hours or as soon as possible after knowledge of the information.

Depending on the nature and seriousness of the AE, Santen may request additional documentation, for example, copies of the ophthalmic and medical record of the subject as well as results of laboratory tests. If the subject was hospitalized, the site should summarize the hospital discharge summary and provide to Santen upon request.

#### 11.1.2.2. Expedited Reporting of Serious Adverse Events

Santen (or designee) will provide the Principal Investigator with a reporting cover letter and an anonymized MedWatch 3500A for expedited reporting of SAEs to the IRB or IEC. The Principal Investigator is responsible for receiving and reviewing expedited safety reports, submitting expedited safety reports to the IRB or IEC, and maintaining copies of expedited safety reports in the study records.

#### 11.1.3. Events of Special Interest

Events of Special Interest (ESIs) are events that may require special attention for the purposes of on-going patient safety review during this study. The following are considered ESIs and should be reported on the appropriate eCRF with as much information as available <u>within 24 hours of knowledge of the event</u>:

- Study medication administration error Study medication administration errors determined to be significant by the Clinical Investigator will be reported and evaluated as ESIs. Examples of study medication administration errors may include, but are not limited to: overdose of study medication and administration of study medication from an incorrect kit.
- **Pregnancy** There are no controlled data with the investigational product in human pregnancy. It is required that women of childbearing potential use effective contraception during the study and recommended for 12 weeks after the completion of the study. Any pregnancy occurring during study treatment should be reported and the subject removed from the study. The subject should be followed until the end of pregnancy or until the end of the study, whichever is longer.
- Ocular telangiectasia and bleeding There is no data showing that the investigational product is related to these events. However, these are seen in the Osler-Weber-Rendu (OWR) syndrome, a genetic condition that causes endoglin dysfunction. DE-122 binds to and suppresses human endoglin, thus information about the ocular manifestations of OWR are of value in predicting possible ocular adverse following IVT injection of DE-122. Any ocular telangiectasia or bleeding (both extra and intraocular) occurring during study treatment should be reported and the subject followed until the end of the study or resolution of the event.

#### 11.1.4. Follow-up of Adverse Events

All reported AEs at study exit will be followed by the Clinical Investigator (or his/her designee) until the event is resolved or determined to be irreversible, chronic, or stable.

In addition, on a case-by-case basis, Santen (or designee) may request follow up beyond the end of the study.

If the Santen Pharmacovigilance Department requests follow-up on an individual SAE or designated ESI, site response to follow-up requests should be faxed to Santen Pharmacovigilance: 415-276-5882 (fax) or drugsafety@santeninc.com.

## 11.1.5. Manual Back-Up Reporting Procedures

This study is utilizing an electronic data capture (EDC) system for data collection. In the event that the EDC system is unavailable for electronic reporting, the manual back-up reporting procedures below should be followed.

- Complete an AE and SAE form.
- Attach a fax cover sheet with your contact information and address to Santen Pharmacovigilance.
- Fax the cover sheet and the AE and SAE form to Santen Pharmacovigilance at

When the EDC system becomes available, update the EDC system with all previously reported information.

# 11.2. Safety Parameters

The safety assessments will include adverse events (AEs), BCVA, slit-lamp biomicroscopy, indirect ophthalmoscopy, intraocular pressure (IOP), serum chemistry, hematology, urinalysis, vital signs, physical exam, fundus photography, fluorescein angiography, EKG, pregnancy.

#### 11.2.1. Physical Examination

A full body systematic physical exam will be conducted by the Clinical Investigator or an external internist during Screening (Day -7 to Day -1) and Visit 8/Exit (Day 90±3).

## 11.2.2. Electrocardiogram (EKG)

EKGs will be performed at Screening (Day -7 to Day -1), Visit 3 (Day 8±1), Visit 5 (Day 30±2) and at Visit 8/Exit (Day 90±3). The Clinical Investigator will review the EKG report for abnormalities.

## 11.2.3. Vital Signs

Blood pressure and heart rate will be measured at each visit using an automated or manual blood pressure monitor. Systolic and diastolic blood pressures will be recorded in millimeters of mercury (mmHg), and heart rate will be recorded in beats per minute (bpm).

#### 11.2.4. Best Corrected Visual Acuity

The BCVA will be recorded using the ETDRS chart and total number of letters at 4 meters and 1 meter will be recorded at each visit. If a subject could not read ETDRS chart, Finger Counts, Hand Motion, Light Perception, or No Light Perception will be recorded.

#### 11.2.5. Slit-lamp Biomicroscopy

Slit-lamp biomicroscopy will be performed at each visit. On the visit of DE-122 or anti-VEGF injection, a biomicroscopy examination will be performed prior to DE-122 or anti-VEGF injection and a second one within 30 minutes after injection.

#### 11.2.6. Intraocular Pressure

IOP will be measured by applanation tonometry and reported in millimeters of mercury (mmHg) at each study visit. On the visit of DE-122 or anti-VEGF injection, IOP will be measured before DE-122 or anti-VEGF injection and 40 ( $\pm$ 10) minutes after injection. If post-injection IOP is increased  $\geq$  10 mmHg from pre-injection IOP, the IOP will be measured again 60 ( $\pm$ 10) minutes following injection. If there is an increase of  $\geq$  10 mmHg at 60 ( $\pm$ 10) minutes post-injection compared to pre-injection IOP, the subject will be prescribed a topical IOP-lowering medication until he or she returns for follow-up per the Clinical Investigator's discretion (an unscheduled visit may apply), and the IOP increase of  $\geq$  10 mmHg shall be reported as an AE.

#### 11.2.7. Indirect Ophthalmoscopy

Indirect ophthalmoscopy will be performed at each visit. On the visit of DE-122 or anti-VEGF injection, an ophthalmoscopy examination will be performed prior to DE-122 or anti-VEGF injection and a second one within 30 minutes after injection.

## 11.2.8. Urine Pregnancy Test

A urine pregnancy test will be conducted at Visit 5 (Day 30±2) and Visit 7 (Day 60±3) for all women of childbearing potential. It should be conducted prior to anti-VEGF IVT injection.

## 11.2.9. Serum Pregnancy Test

A serum pregnancy test will be conducted at Screening (Day -7 to Day -1) and Visit 8/Exit (Day 90±3) for all women of childbearing potential.

#### 11.2.10. Serum Chemistry, Hematology and Urinalysis

A fasting blood sample and urine sample will be taken at Screening (Day -7 to Day -1), Visit 3 (Day 8±1), Visit 5 (Day 30±2), and Visit 8/Exit (Day 90±3).

## 11.2.11. Fundus Photography

Digital color fundus photography will be taken at Screening (Day -7 to Day -1), Visit 5 (Day 30±2), Visit 7 (Day 60±3) and Visit 8/Exit (Day 90±3) in both eyes. At Visit 5 (Day 30±2), it will be performed prior to anti-VEGF injection. Required fields to be captured are: Nasal to macula (The image is centered on the optic nerve), Posterior pole (The image is centered on the macula).

#### 11.2.12. Fluorescein Angiography

Fundus fluorescein angiography will be taken at Screening (Day -7 to Day -1), Visit 5 (Day 30±2), Visit 7 (Day 60±3) and Visit 8/Exit (Day 90±3) in both eyes. At Visit 5 (Day 30±2), it will be performed prior to anti-VEGF injection. Required fields to be captured are: Nasal to macula (The image is centered on the optic nerve), Posterior pole (The image is centered on the macula).

#### 11.2.13. Adverse Events

AEs will be elicited from the subjects starting at the Screening (Day -7 to Day -1) through Visit 8/Exit (Day 90±3). The information will include at least a description of the event, whether or not it is serious, onset and duration, frequency, severity, relation to DE-122, relation to injection procedure, location (OD, OS, OU or NA), action taken and outcome. Prior to evaluating the incidences, all AEs will be coded using the Medical Dictionary for Regulatory Activities (MedDRA, 2013). Ocular and non-ocular AEs will be summarized separately. See Section 11.1 for complete information regarding AE reporting.

## 12. ASSESSMENT OF BIOACTIVITY

Measures to assess bioactivity include subretinal fluid and macular volume. The effects of DE-122 on resolution of subretinal fluid will be assessed using the change in CST and the macular volume based on SD-OCT.

SD-OCT will be performed for both eyes at each visit. CST, an average of central subfield thickness, will be recorded. In addition, macular volume will be determined.

#### 13. OTHER ASSESSMENTS

# **13.1.** Demographics and Baseline Characteristics

Subject demographics include age, race, sex, and ethnicity. Baseline characteristics include medical history, prior medications, and baseline results of physical exam, EKG, vital signs, BCVA, slit-lamp biomicroscopy, IOP, indirect ophthalmoscopy, SD-OCT, pregnancy test, laboratory tests (hematology, chemistry, and urinalysis), fundus photography and fluorescein angiography. For assessments performed multiple times before the injection of IVT DE-122, the last pre-injection value will be used as the baseline value.

# 13.2. Immunogenicity

ADA titer will be measured in serum samples collected at Visit 1 (Day 1) and Visit 5 (Day 30±2).

#### 13.3. Biomarker

For the biomarker finding, serum samples will be collected according examination schedule from the subjects in Cohorts 3 and 4, and measured for levels of endoglin-related proteins. The remaining serum samples will be stored for future exploratory research to identify possible other biomarkers associated with the study drug(s) and/or ophthalmologic disease conditions.

#### 13.4. Other Assessments

Other assessments include concomitant medications and exposure to study drug.

#### 14. STATISTICAL METHODS

#### 14.1. General Considerations

All study parameters will be listed and a selected list of parameters will be summarized descriptively by dose level and overall. The descriptive statistics will include number of observations (n), mean, standard deviation, minimum, and maximum for continuous parameter and frequency (n) and percent (%) for categorical parameters.

Details about the statistical analyses for this study will be provided in the statistical analysis plan (SAP).

All data manipulations and descriptive summaries will be implemented using SAS®, Version 9.1.3 or later

#### 14.1.1. Study Endpoints

Safety:

• Incidence and severity of adverse events (AEs), slit-lamp biomicroscopy, indirect ophthalmoscopy, BCVA, IOP, fundus photography, fluorescein angiography, serum chemistry, hematology, urinalysis, vital signs, physical exam, EKG and pregnancy

#### Bioactivity:

• Change in CST and macular volume based on SD-OCT at each visit post DE-122 treatment

#### 14.1.2. Sample Size

Approximately twelve subjects (2 or 3 subjects in Cohort 1; 3 subjects in Cohorts 2, 3, and 4) with refractory exudative age related macular degeneration will be enrolled at 5 sites. The final number of subjects enrolled may be adjusted based on the presence of dose limiting toxicities. This sample size is not planned based on statistical considerations.

## 14.1.3. Statistical Hypotheses and Level of Significance

No statistical hypothesis is defined for this study.

#### 14.1.4. Randomization

This is an open-label, non-randomized study.

#### **14.1.5.** Study Eye

The study eye is defined as the eye with worse vision. If both eyes have the same vision, the right eye (OD) should be determined as the study eye.

## 14.2. Study Populations

The following study populations are defined for analysis: Intention-to-treat (ITT) and Safety.

**ITT Population**: The ITT population will include all subjects in the study. It will be the primary study population for bioactivity analyses, where subjects are grouped by planned dose level unless specified otherwise.

**Safety Population**: The Safety population will include all subjects who receive the injection of IVT DE-122. It will be the study population for safety analyses performed with subjects as treated.

# 14.3. Handling of Missing Values

For safety measures, missing scores will not be imputed for data summaries.

Completely or partially missing onset and resolution dates for AEs and completely or partially missing start and end dates of concomitant medications will be imputed in a conservative fashion that will be detailed in the SAP.

For Bioactivity endpoints, missing post-injection values will be imputed using the last-observation-carried-forward (LOCF) approach.

# 14.5. Demographics and Baseline Characteristics

Age, sex, race, ethnicity, and baseline assessments will be summarized descriptively by dose level.

Subjects with abnormal medical history will be tabulated by treatment arm and body system.

Subjects using any prior medications will be tabulated by dose level, Anatomical Therapeutic Chemical levels, and preferred term specified in the World Health Organization Drug Dictionary Enhanced (World Health Organization Drug Dictionary Enhanced, 2011).

# 14.6. Bioactivity Analyses

Changes from baseline in BCVA, retinal thickness (CST), and macular volume will be summarized descriptively by dose level of DE-122. Change in retinal thickness after anti-VEGF injection will also be provided.

# 14.7. Safety Analysis

All safety outcome measures will be summarized descriptively for the Safety Population. The safety outcome measures include adverse events (AEs), BCVA, slit-lamp biomicroscopy, indirect ophthalmoscopy, intraocular pressure (IOP), serum chemistry, hematology, urinalysis, vital signs, physical exam, fundus photography, fluorescein angiography, EKG and pregnancy.

AEs will be coded using the Medical Dictionary for Regulatory Activities (MedDRA).

Subjects with any AEs will be tabulated by system organ classification and preferred term specified in the MedDRA. Similarly, subjects with any ocular and non-ocular AEs and ESIs will be tabulated separately. AEs, ocular and non-ocular, as well as ESIs will also be summarized by relationship to treatment and maximum severity. In addition, SAEs and discontinuations due to AEs will be summarized.

Ocular safety outcome measures will be summarized using descriptive statistics.

# 14.8. Other Analysis

# 14.8.1. Immunogenicity Analysis

To assess immunogenicity, the incidence of DE-122 antibody development in each cohort will be summarized by frequency counts and percentages.

# 14.8.2. Biomarker Analysis

Changes from baseline in levels of biomarkers will be summarized descriptively by dose level of DE-122.

## 15. DIRECT ACCESS TO SOURCE DATA/DOCUMENTS

The Principal Investigator will allow representatives of Santen's monitoring team (or designee), the governing institutional review board (IRB), the FDA, and other applicable regulatory agencies to inspect all study records, eCRFs, recruitment materials and corresponding portions of the subject's medical records at regular intervals throughout the study. These inspections are for the purpose of verifying adherence to the protocol, completeness, and exactness of the data being entered onto the eCRF, and compliance with the FDA or other regulatory agency regulations.

# 15.1. Study Monitoring

Before an investigational site can enter a subject into the study, a representative of Santen (or designee) will evaluate the investigational study site to:

- Determine the adequacy of the study facilities.
- Review with the Principal Investigator(s) and authorized study staff their responsibilities with regard to protocol procedures adherence, and the responsibilities of Santen (or designee).

During the study, Santen (or designee) will have regular contact with the investigational site, for the following:

- Provide information and support to the Principal Investigator(s).
- Confirm that facilities remain acceptable.
- Assess adherence to the protocol and GCP.
- Perform investigational product accountability checks and quality control procedures.
- Ensure the on-going implementation of accurate data entry in the eCRF.
- Perform source data verification, including a comparison of the data in the eCRFs with the subject's medical records and other records relevant to the study. This will require direct access to all original records for each subject (e.g., clinic charts).
- Record and report any protocol deviations not previously sent to Santen.
- Confirm AEs and SAEs have been properly documented on eCRFs and confirm any SAEs have been forwarded to Santen and those SAEs that met criteria for reporting have been forwarded to the IRB or Independent Ethics Committee (IEC).

Santen (or designee) may remotely access the eCRFs at any time during the study for centralized monitoring. Santen (or designee) will be available between visits if authorized study staff needs study related information or support.

# 15.2. Audits and Inspections

The Principal Investigator will allow Santen (or designee), the governing IRB or IEC, and applicable regulatory agencies to audit and inspect any aspect of the study, including all study records, eCRFs, recruitment materials, and corresponding portions of the subject's charts and

medical records at any time during the study. These study records must be retained at the study site and made available for audits and inspections. The purpose of these audits and inspections is to verify adherence to the protocol, completeness and accuracy of the eCRF data, and compliance with Good Clinical Practice (GCP) guidelines and applicable regulatory requirements.

The Principal Investigator or authorized study staff will notify Santen (or designee) should the site be audited or inspected by the governing IRB or IEC, and applicable regulatory agencies. Santen (or designee) will also notify the investigational site of any known pending site audits or inspections planned by Santen (or designee), governing IRB or IEC and regulatory agencies.

#### 15.3. Institutional Review Board

The Principal Investigator must obtain IRB approval for the investigation. Initial IRB approval, and all materials approved by the IRB for this study including the subject consent form and recruitment materials must be maintained by the Principal Investigator and made available for inspection.

## 16. QUALITY CONTROL AND QUALITY ASSURANCE

# 16.1. Quality Control

Santen (or designee) will provide instructional material to the study sites, as appropriate; including but not limited to instruction on the protocol, the completion of eCRFs, and study procedures. Santen (or designee) will communicate regularly with site personnel via mail, email, telephone, and/or fax; and make periodic visits to the study site. During those visits, Santen (or designee) will perform source data verification with the subject's medical records and other records relevant to the study. Upon receiving the eCRFs, Santen (or designee) will review and evaluate eCRF data and use standard system edits and may use centralized monitoring to detect errors in data collection.

# 16.2. Quality Assurance

Santen (or designee) may conduct a quality assurance audit at any time.

## 17. ETHICS

#### 17.1. Ethics Review

The final study protocol and the final version of the ICF, and other study related material, as appropriate, must be approved or given a favorable opinion in writing by an IRB or IEC as appropriate. The Principal Investigator must submit written approval to Santen (or designee) before study initiation. See Section 21.1 Appendix A for a list of obligations of Investigators.

The Principal Investigator is responsible for informing the IRB or IEC of any amendment to the protocol in accordance with local regulations and guidelines. In addition, the IRB or IEC must approve all advertising used to recruit subjects for the study. The protocol must be re-approved by the IRB or IEC upon receipt of amendments and at least annually.

The Principal Investigator is also responsible for providing the IRB or IEC with progress reports and notifications of any reportable serious adverse drug reactions from the investigational product.

## 17.2. Ethical Conduct of the Study

This study will be conducted in compliance with IRB or IEC, and regulatory requirements. This study will also be conducted in compliance with the protocol, GCP guidelines, International Conference on Harmonization (ICH) guidelines, the Declaration of Helsinki, and Health Insurance Portability and Accountability Act of 1996 (HIPAA).

#### 17.3. Written Informed Consent

The Principal Investigator at each center will ensure that the subject is given full and adequate oral and written information about the nature, purpose, possible risk and possible benefit of the study. Subjects must also be notified that they are free to withdraw from the study at any time. Subjects should be given the opportunity to ask questions and allowed time to consider the information provided. Before participating in any study-related activity, voluntary informed consent must be documented by the use of a written ICF approved by the IRB or IEC and signed and dated by the subject or the subject's legally authorized representative at the time of consent. The original signed and dated ICF will be retained with the study records, and a copy of the signed ICF will be given to the subject or the subject's legally authorized representative.

#### 18. DATA HANDLING AND RECORDKEEPING

# **18.1.** Inspection of Records

The Principal Investigator will allow Santen (or designee), the governing IRB or IEC and applicable regulatory agencies to inspect any aspect of the study, including all study records, eCRFs, recruitment materials and corresponding portions of the subject's charts and medical records at any time during the study. The purpose of these inspections is to verify adherence to the protocol, completeness and accuracy of the eCRF data, and compliance with GCP guidelines and applicable regulatory requirements.

#### 18.2. Retention of Records

All records relating to the conduct of this study are to be retained by the Principal Investigator until notified by Santen (or designee) that the records may be destroyed.

#### 18.2.1. Source Documents

The Principal Investigator must maintain detailed source documents on all study subjects who provide informed consent. Source documents include subject medical records, hospital charts, study files, as well as the results of diagnostic tests (e.g., laboratory tests).

The following minimum information should be entered into the subject's medical record:

- The date the subject was enrolled and the subject number
- The study protocol number and the name of Santen Inc.
- The date that informed consent was obtained
- Evidence that the subject meets study eligibility requirements (e.g., medical history, study procedures and/or evaluations)
- The dates of all study-related subject visits
- Evidence that required procedures and/or evaluations were completed
- Use of any concomitant medications
- Documentation of study drug accountability
- Occurrence and status of any AEs
- The date the subject exited the study and a notation as to whether the subject completed or terminated early from the study, including the reason for early termination

#### 18.2.2. Data Collection

The Principal Investigator must maintain detailed records on all subjects who provide informed consent. Data for screened and enrolled subjects will be entered into eCRFs. Review of the eCRFs will be completed remotely by Santen (or designee). At designated intervals, a study monitor will perform source data verification on site. During those visits, Santen (or designee) will monitor the subject data recorded in the eCRF against source documents at the study site. Santen (or designee) will review and evaluate eCRF data and use standard system edits, and may use centralized monitoring evaluations, to detect errors in data collection. At the end of the study, a copy of the completed eCRFs will be sent to the site to be maintained as study records.

#### 19. PUBLICATION POLICY

The existence of this clinical study is confidential, and it should not be discussed with persons outside of the study. Additionally, the information in this document and regarding this study contains trade secrets and commercially sensitive information that is confidential and may not be disclosed unless such disclosure is required by federal or state law or regulations. Subject to the foregoing, this information may be disclosed only to those persons involved in the study who have a need to know, but all such persons must be instructed not to further disseminate this information to others. These restrictions of disclosure will apply equally to all future information supplied that is indicated as confidential. Information pertaining to this study will be published on www.clinicaltrials.gov as required by the Food and Drug Administration (FDA).

The data generated by this clinical study are the property of Santen and should not be disclosed without the prior written permission of Santen. These data may be used by Santen now and in the future for presentation or publication at Santen's discretion or for submission to governmental regulatory agencies. Santen reserves the right of prior review of any publication or presentation of data from this study.

In signing this protocol, the Principal Investigator agrees to the release of the data from this study and acknowledges the above publication policy.

#### 20. REFERENCES

- 1. Barbara, N., Wrana, J., Letarte, M. (1999). Endoglin Is an Accessory Protein That Interacts with the Signaling Receptor Complex of Multiple Members of the Transforming Growth Factor-b Superfamily. The Journal of Biological Chemistry 274(2):584-94.
- 2. Gordon, M., Kass, M. (2001). Ocular Hypertension Treatment Study (OHTS), Manual of Procedures, Version 3.0. National Technical Information Service.
- 3. Guo, B., Slevin, M., Li, C., Parameshwar, S., Liu, D., Kumar, P., Bernabeu, C., Kumar, S. (2004). CD105 Inhibits Transforming Growth Factor-β-Smad3 Signalling. Anticancer Research 24(3a):1337-45.
- Heier, J., Brown, D., Chong, V., Korobelnik, J., Kaiser, P., Nguyen, Q., Kirchhof, B., Ho, A., Ogura, Y., Yancopoulos, G., Stahl, N., Vitti, R., Berliner, A., Soo, Y., Anderesi, M., Groetzbach, G., Sommerauer, B., Sandbrink, R., Simader, C., Schmidt-Erfurth, U. (2012). Intravitreal Aflibercept (VEGF Trap-Eye) in Wet Age-related Macular Degeneration. Ophthalmology 119(12):2537-48.
- 5. Kane, F., Campochiaro, P. (2008). Choroidal Neovascularization. In: Lim J, editor. Age-Related Macular Degeneration. 2nd ed. Chapter 5; p. 87-95.
- 6. Lebrin, F., Goumans, M., Jonker, L., Carvalho, R., Valdimarsdottir, G., Thorikay, M., Mummery, C., Arthur, H., ten Dijke, P. (2004). Endoglin promotes endothelial cell proliferation and TGF-b/ALK1 signal transduction. The EMBO Journal 23(20):4018-28.
- 7. Li, C., Issa, R., Kumar, P., Hampson, I., Lopez-Novoa, J., Bernabeu, C., Kumar, S. (2003). CD105 prevents apoptosis in hypoxic endothelial cells. Journal of Cell Science 116(13):2677-85.
- 8. Lim, J., Tsong, J. (2008). Exudative (Neovascular) Age-Related Macular Degeneration. In: Lim J, editor. Age-Related Macular Degeneration. 2nd ed. Chapter 8; p. 125-57.
- 9. MedDRA MSSO, Medical Dictionary for Regulatory Activities, Version 16.1. Available from http://www.meddra.org/
- 10. Nolan-Stevaux, O., Zhong, W., Culp, S., Shaffer, K., Hoover, J., Wickramasinghe, D., Ruefli-Brasse, A. (2012). Endoglin Requirement for BMP9 Signaling in Endothelial Cells Reveals New Mechanism of Action for Selective Anti-Endoglin Antibodies. PLoS ONE 7(12):1-12.
- 11. Nussenblatt, R., Palestine, A., Chan, C., Roberge, F. (1985). Standardization of Vitreal Inflammatory Activity in Intermediate and Posterior Uveitis. Ophthalmology 92(4):467-71.

- 12. Park, S., Lee, Y., Seki, T., Hong, K., Fliess, N., Jiang, Z., Park, A., Wu, X., Kaartinen, V., Roman, B., Oh, S. (2008). ALK5- and TGFBR2-independent role of ALK1 in the pathogenesis of hereditary hemorrhagic telangiectasia type 2. Blood 111(2):633-42.
- 13. Sun Working Group. (2005). PERSPECTIVES Standardization of Uveitis Nomenclature or Reporting Clinical Data. Results of the First International Workshop. American Journal of Ophthalmology 140(3):509-16.
- 14. U.S.Department of Health and Human Services, National Institutes of Health. (01 Aug 2004). The Seventh Report of the Joint National Committee on Prevention, Detection, Evaluation, and Treatment of High Blood Pressure.
- 15. Warrington, K., Hillarby, M., Li, C., Letarte, M., Kumar, S. (2005). Functional Role of CD105 in TGF-b1 Signalling in Murine and Human Endothelial Cells. Anticancer Research 25(3B):1851-64.
- 16. World Health Organization Drug Dictionary Enhanced. World Health Organization Drug Dictionary Enhanced (WHO-DDE), September 2011 Version. Available from <a href="http://www.umc-products.com/DynPage.aspx?id=73588&mn1=1107&mn2=1139">http://www.umc-products.com/DynPage.aspx?id=73588&mn1=1107&mn2=1139</a>
- 17. Yasukawa, T., Kimura, H., Tabata, Y., Miyamoto, H., Honda, Y., Ikada, Y., Ogura, Y. (2000). Active drug targeting with immunoconjugates to choroidal neovascularization. Current Eye Research 21(6):952-61.

#### 21. APPENDICES

# 21.1. Appendix A - Obligations of Investigators

In summary, the Clinical Investigator has agreed to the following obligations:

- Obtaining informed consent from every subject prior to the subject's participation in any study related activity and maintaining records of consent as part of the study records.
- Obtaining approval from the IRB before involving any subject in any study related activity; submitting verification of the approval to the Sponsor; submitting periodic progress reports (at least annually) and final report to IRB and to the Sponsor.
- Approving the protocol and conducting the study according to the protocol and applicable regulations; informing the Sponsor of all deviations from the protocol.
- Informing the IRB of all protocol amendments/modifications; sending the Sponsor a copy of the letter from the IRB approving the amendment/modification.
- Reporting to the Sponsor and the IRB any adverse experiences that occur in the course of the investigation, this includes Serious Adverse Events within 24 hours.
- Keeping careful and accurate records of all clinical study data (study records must be
  considerably more exact and complete than those kept in ordinary medical practice);
  maintaining records of all materials submitted to the IRB and of all action by the IRB
  regarding the study.
- Making study records available for inspection by the Sponsor and representatives of the Food and Drug Administration and other regulatory agencies; keeping records until notified by the Sponsor that they may be destroyed.
- Maintaining proper control and documentation of all test and control articles.
- Submitting the following records and reporting to the Sponsor (Section 21.1).

## I. Prior to the Beginning of the Study

- A signed Form FDA-1572, Statement of Investigator.
- A current curriculum vitae (CV) if not submitted to Santen previously or if updated.
- CVs for all sub-Investigators listed on the 1572.
- A letter from the IRB indicating that the protocol was approved, including the name and address of the IRB.
- A copy of the consent form approved by IRB.
- A list of current members of the IRB.

## **II.** While the Study Is in Progress

- Acknowledgment of receipt of the test and control articles; documentation of disposition of all test and control articles.
- Original Case Report Forms for each subject enrolled in the study.
- Information regarding all deviations from the protocol.
- Information regarding all adverse medical events occurring to a subject while enrolled in the study.
- Annual progress report (if study is ongoing for more than one year). Letter from the IRB indicating approval of the annual progress report.

## III. Once the Study Is Completed

- Disposition of all used and/or unused test and control articles, as well as documentation of all drug accountability.
- A final study report.

# 21.2. Appendix B - Elements of Informed Consent

#### I. Elements of Informed Consent

The following information must be provided to each subject in obtaining informed consent. If written consent is being obtained, the subject (or subject's legal representative) should be provided with a copy of the signed written ICF.

- 1. State that the study involves RESEARCH.
  - A. Explain the PURPOSE of the research.
  - B. Trial treatments and the probability for random assignment to each treatment.
  - C. State the expected DURATION of the subject's participation.
  - D. Describe the PROCEDURES to be followed.
  - E. Identify any EXPERIMENTAL procedures.
- 2. Describe any reasonably foreseeable RISKS OR DISCOMFORTS to the subject.
- 3. Describe any BENEFITS to the subject and responsibility for the subject or to others that may reasonably be expected from the research.
- 4. Note appropriate ALTERNATIVE procedures or courses of treatment, if any, that might be advantageous to the subject.
- 5. A. Describe the extent, if any, to which CONFIDENTIALITY of records identifying the subject will be maintained.
  - B. Note that the FDA MAY INSPECT the records.
- 6. For research involving more than minimal risk, explain if any COMPENSATION or medical treatments are available should injury occur. If so, explain (a) what they consist of, OR (b) where further information may be obtained.
- 7. A. Tell whom to contact for ANSWERS to pertinent questions about (a) the research, and (b) research subjects' rights.
  - B. Tell whom to contact in the event of a research-related INJURY to the subject.
- 8. State that:
  - A. Participation is VOLUNTARY.
  - B. Refusal to participate will involve NO PENALTY or loss of benefits to which the subject is otherwise entitled
  - C. The subject MAY DISCONTINUE participation at any time without penalty or loss of benefits to which the subject is otherwise entitled.

#### II. Additional Elements of Informed Consent

When appropriate, one or more of the following elements of information shall also be provided to each subject:

- 1. A statement that particular treatment or procedure may involve risks to the subject (or to the embryo or fetus, if the subject is or may become pregnant) which are currently unforeseeable.
- 2. Anticipated circumstances under which the subject's participation may be terminated by the Investigator without regard to the subject's consent.
- 3. Any additional costs to the subject that may result from participation in the research.
- 4. The consequences of a subject's decision to withdraw from the research and procedures for orderly termination of participation by the subject.
- 5. A statement that significant new findings developed during the course of the research, which may relate to the subject's willingness to continue participation, will be provided to the subject.
- 6. The approximate number of subjects involved in the study.

The informed consent requirements in this protocol are not intended to preempt any applicable Federal, State, or local laws which require additional information to be disclosed for informed consent to be legally effective.

Nothing in this protocol is intended to limit the authority of a physician to provide emergency medical care to the extent the physician is permitted to do so under applicable Federal, State, or local law.

REFERENCE: 21 CFR Part 50.25 – PROTECTION OF HUMAN SUBJECTS, Elements of Informed Consent.

# 21.3. Appendix C - Declaration of Helsinki WMA Declaration of Helsinki - Ethical Principles for Medical Research Involving Human Subjects

Adopted by the 18th WMA General Assembly, Helsinki, Finland, June 1964 and amended by the:

29th WMA General Assembly, Tokyo, Japan, October 1975
35th WMA General Assembly, Venice, Italy, October 1983
41st WMA General Assembly, Hong Kong, September 1989
48th WMA General Assembly, Somerset West, Republic of South Africa, October 1996
52nd WMA General Assembly, Edinburgh, Scotland, October 2000
53rd WMA General Assembly, Washington DC, USA, October 2002 (Note of Clarification added)
55th WMA General Assembly, Tokyo, Japan, October 2004 (Note of Clarification added)

59th WMA General Assembly, Seoul, Republic of Korea, October 2008 64th WMA General Assembly, Fortaleza, Brazil, October 2013

#### **Preamble**

1. The World Medical Association (WMA) has developed the Declaration of Helsinki as a statement of ethical principles for medical research involving human subjects, including research on identifiable human material and data.

The Declaration is intended to be read as a whole and each of its constituent paragraphs should be applied with consideration of all other relevant paragraphs.

2. Consistent with the mandate of the WMA, the Declaration is addressed primarily to physicians. The WMA encourages others who are involved in medical research involving human subjects to adopt these principles.

#### **General Principles**

- 3. The Declaration of Geneva of the WMA binds the physician with the words, "The health of my patient will be my first consideration," and the International Code of Medical Ethics declares that, "A physician shall act in the patient's best interest when providing medical care."
- 4. It is the duty of the physician to promote and safeguard the health, well-being and rights of patients, including those who are involved in medical research. The physician's knowledge and conscience are dedicated to the fulfilment of this duty.
- 5. Medical progress is based on research that ultimately must include studies involving human subjects.
- 6. The primary purpose of medical research involving human subjects is to understand the causes, development and effects of diseases and improve preventive, diagnostic and therapeutic interventions (methods, procedures and treatments). Even the best proven interventions must be evaluated continually through research for their safety, effectiveness, efficiency, accessibility and quality.
- 7. Medical research is subject to ethical standards that promote and ensure respect for all human subjects and protect their health and rights.

- 8. While the primary purpose of medical research is to generate new knowledge, this goal can never take precedence over the rights and interests of individual research subjects.
- 9. It is the duty of physicians who are involved in medical research to protect the life, health, dignity, integrity, right to self-determination, privacy, and confidentiality of personal information of research subjects. The responsibility for the protection of research subjects must always rest with the physician or other health care professionals and never with the research subjects, even though they have given consent.
- 10. Physicians must consider the ethical, legal and regulatory norms and standards for research involving human subjects in their own countries as well as applicable international norms and standards. No national or international ethical, legal or regulatory requirement should reduce or eliminate any of the protections for research subjects set forth in this Declaration.
- 11. Medical research should be conducted in a manner that minimizes possible harm to the environment.
- 12. Medical research involving human subjects must be conducted only by individuals with the appropriate ethics and scientific education, training and qualifications. Research on patients or healthy volunteers requires the supervision of a competent and appropriately qualified physician or other health care professional.
- 13. Groups that are underrepresented in medical research should be provided appropriate access to participation in research.
- 14. Physicians who combine medical research with medical care should involve their patients in research only to the extent that this is justified by its potential preventive, diagnostic or therapeutic value and if the physician has good reason to believe that participation in the research study will not adversely affect the health of the patients who serve as research subjects.
- 15. Appropriate compensation and treatment for subjects who are harmed as a result of participating in research must be ensured.

#### Risks, Burdens and Benefits

16. In medical practice and in medical research, most interventions involve risks and burdens.

Medical research involving human subjects may only be conducted if the importance of the objective outweighs the risks and burdens to the research subjects.

17. All medical research involving human subjects must be preceded by careful assessment of predictable risks and burdens to the individuals and groups involved in the research in comparison with foreseeable benefits to them and to other individuals or groups affected by the condition under investigation.

Measures to minimize the risks must be implemented. The risks must be continuously monitored, assessed and documented by the researcher.

18. Physicians may not be involved in a research study involving human subjects unless they are confident that the risks have been adequately assessed and can be satisfactorily managed.

When the risks are found to outweigh the potential benefits or when there is conclusive proof of definitive outcomes, physicians must assess whether to continue, modify or immediately stop the study.

#### **Vulnerable Groups and Individuals**

19. Some groups and individuals are particularly vulnerable and may have an increased likelihood of being wronged or of incurring additional harm.

All vulnerable groups and individuals should receive specifically considered protection.

20. Medical research with a vulnerable group is only justified if the research is responsive to the health needs or priorities of this group and the research cannot be carried out in a non-vulnerable group. In addition, this group should stand to benefit from the knowledge, practices or interventions that result from the research.

## Scientific Requirements and Research Protocols

- 21. Medical research involving human subjects must conform to generally accepted scientific principles, be based on a thorough knowledge of the scientific literature, other relevant sources of information, and adequate laboratory and, as appropriate, animal experimentation. The welfare of animals used for research must be respected.
- 22. The design and performance of each research study involving human subjects must be clearly described and justified in a research protocol.

The protocol should contain a statement of the ethical considerations involved and should indicate how the principles in this Declaration have been addressed. The protocol should include information regarding funding, sponsors, institutional affiliations, potential conflicts of interest, incentives for subjects and information regarding provisions for treating and/or compensating subjects who are harmed as a consequence of participation in the research study.

In clinical trials, the protocol must also describe appropriate arrangements for post-trial provisions.

#### **Research Ethics Committees**

23. The research protocol must be submitted for consideration, comment, guidance and approval to the concerned research ethics committee before the study begins. This committee must be transparent in its functioning, must be independent of the researcher, the sponsor and any other undue influence and must be duly qualified. It must take into consideration the laws and regulations of the country or countries in which the research is to be performed as well as applicable international norms and standards but these must not be allowed to reduce or eliminate any of the protections for research subjects set forth in this Declaration.

The committee must have the right to monitor ongoing studies. The researcher must provide monitoring information to the committee, especially information about any serious adverse events. No amendment to the protocol may be made without consideration and approval by the committee. After the end of the study, the researchers must submit a final report to the committee containing a summary of the study's findings and conclusions.

#### **Privacy and Confidentiality**

24. Every precaution must be taken to protect the privacy of research subjects and the confidentiality of their personal information.

## **Informed Consent**

- 25. Participation by individuals capable of giving informed consent as subjects in medical research must be voluntary. Although it may be appropriate to consult family members or community leaders, no individual capable of giving informed consent may be enrolled in a research study unless he or she freely agrees.
- 26. In medical research involving human subjects capable of giving informed consent, each potential subject must be adequately informed of the aims, methods, sources of funding, any possible conflicts of interest, institutional affiliations of the researcher, the anticipated benefits and potential risks of the study and the discomfort it may entail, post-study provisions and any other relevant aspects of the study. The potential subject must be informed of the right to refuse to participate in the study or to withdraw consent to participate at any time without reprisal. Special attention should be given to the specific information needs of individual potential subjects as well as to the methods used to deliver the information.

After ensuring that the potential subject has understood the information, the physician or another appropriately qualified individual must then seek the potential subject's freely-given informed consent, preferably in writing. If the consent cannot be expressed in writing, the non-written consent must be formally documented and witnessed.

All medical research subjects should be given the option of being informed about the general outcome and results of the study.

- 27. When seeking informed consent for participation in a research study the physician must be particularly cautious if the potential subject is in a dependent relationship with the physician or may consent under duress. In such situations the informed consent must be sought by an appropriately qualified individual who is completely independent of this relationship.
- 28. For a potential research subject who is incapable of giving informed consent, the physician must seek informed consent from the legally authorized representative. These individuals must not be included in a research study that has no likelihood of benefit for them unless it is intended to promote the health of the group represented by the potential subject, the research cannot instead be performed with persons capable of providing informed consent, and the research entails only minimal risk and minimal burden.
- 29. When a potential research subject who is deemed incapable of giving informed consent is able to give assent to decisions about participation in research, the physician must seek that assent in addition to the consent of the legally authorized representative. The potential subject's dissent should be respected.
- 30. Research involving subjects who are physically or mentally incapable of giving consent, for example, unconscious patients, may be done only if the physical or mental condition that prevents giving informed consent is a necessary characteristic of the research group. In such circumstances the physician must seek informed consent from the legally authorized representative. If no such representative is available and if the research cannot be delayed, the study may proceed without informed consent provided that the specific reasons for involving
subjects with a condition that renders them unable to give informed consent have been stated in the research protocol and the study has been approved by a research ethics committee. Consent to remain in the research must be obtained as soon as possible from the subject or a legally authorized representative.

- 31. The physician must fully inform the patient which aspects of their care are related to the research. The refusal of a patient to participate in a study or the patient's decision to withdraw from the study must never adversely affect the patient-physician relationship.
- 32. For medical research using identifiable human material or data, such as research on material or data contained in biobanks or similar repositories, physicians must seek informed consent for its collection, storage and/or reuse. There may be exceptional situations where consent would be impossible or impracticable to obtain for such research. In such situations the research may be done only after consideration and approval of a research ethics committee.

# **Use of Placebo**

33. The benefits, risks, burdens and effectiveness of a new intervention must be tested against those of the best proven intervention(s), except in the following circumstances:

Where no proven intervention exists, the use of placebo, or no intervention, is acceptable; or

Where for compelling and scientifically sound methodological reasons the use of any intervention less effective than the best proven one, the use of placebo, or no intervention is necessary to determine the efficacy or safety of an intervention

and the patients who receive any intervention less effective than the best proven one, placebo, or no intervention will not be subject to additional risks of serious or irreversible harm as a result of not receiving the best proven intervention.

Extreme care must be taken to avoid abuse of this option.

# **Post-Trial Provisions**

34. In advance of a clinical trial, sponsors, researchers and host country governments should make provisions for post-trial access for all participants who still need an intervention identified as beneficial in the trial. This information must also be disclosed to participants during the informed consent process.

# Research Registration and Publication and Dissemination of Results

- 35. Every research study involving human subjects must be registered in a publicly accessible database before recruitment of the first subject.
- 36. Researchers, authors, sponsors, editors and publishers all have ethical obligations with regard to the publication and dissemination of the results of research. Researchers have a duty to make publicly available the results of their research on human subjects and are accountable for the completeness and accuracy of their reports. All parties should adhere to accepted guidelines for ethical reporting. Negative and inconclusive as well as positive results must be published or otherwise made publicly available. Sources of funding, institutional affiliations and conflicts of interest must be declared in the publication. Reports of research not in accordance with the principles of this Declaration should not be accepted for publication.

# **Unproven Interventions in Clinical Practice**

37. In the treatment of an individual patient, where proven interventions do not exist or other known interventions have been ineffective, the physician, after seeking expert advice, with informed consent from the patient or a legally authorized representative, may use an unproven intervention if in the physician's judgment it offers hope of saving life, re-establishing health or alleviating suffering. This intervention should subsequently be made the object of research, designed to evaluate its safety and efficacy. In all cases, new information must be recorded and, where appropriate, made publicly available.

# 21.4. Appendix D - Procedures for Examinations

# 21.4.1. Demographics/Eligibility, Medical/Surgical History and Concomitant Medication

Demographics/Eligibility, medical/surgical history and concomitant medication will be obtained through subject interviews at Screening (Day -7 to Day -1). Medical history and concomitant medications will be obtained through subject interviews at each visit. CST before the recent anti-VEGF medication received at > 30 days and < 60 days from Visit 1 (Day 1) will be collected as a Medical History.

# 21.4.2. Physical Examination

A full body systematic physical exam will be conducted during Screening (Day -7 to Day -1) and Visit 8/Exit (Day 90±3). Clinical Investigator or an external internist will confirm subject's overall condition noting any abnormalities by a review of the following systems: e.g., head, eyes, ears, nose and throat (HEENT), cardiopulmonary, endocrine, gastrointestinal, musculoskeletal/rheumatic, neurologic/psychiatric, dermatologic, hepatic/renal systems, and other.

The Clinical Investigator will assess subject's overall condition to determine qualification for study entry considering possible class effects of DE-122. Newly noted abnormalities or worsening of previously noted abnormalities found at Study Exit, or at any safety assessment visit, will be assessed as an AE. The Clinical Investigator should use his or her clinical judgment for appropriate treatment and/or medical referral.

# 21.4.3. Vital Signs

Blood pressure and heart rate will be measured at each visit using an automated or manual blood pressure monitor. Systolic and diastolic blood pressures will be recorded in millimeters of mercury (mmHg) and heart rate will be recorded in beats per minute (bpm).

In accordance with the recommendations of the Joint National Committee on Prevention, Detection, Evaluation, and Treatment of High Blood Pressure (U.S.Department of Health and Human Services et al., 2004), the following measurement procedure will be used to measure vital signs:

- Subject should not smoke or ingest caffeine within the 30-minute period immediately before the measurement.
- Subject should be seated quietly in a chair with the back supported, feet on the floor, arm bared, and arm supported at heart level.
- Begin the measurement after at least 5 minutes of rest.
- To ensure an accurate measurement, use an appropriately sized cuff. The cuff bladder should encircle at least 80% of the arm. Many adults need a large cuff.
- Take two (2) systolic/diastolic pressure and heart rate measurements separated by at least 30 seconds. Record each measurement in the subject's source document.

- If the two pressure measurements <u>differ by 5 mmHg or less</u>, then the average of the two becomes the recorded pressure. For example, if the two measurements are 120/90 and 125/95, then 122.5/92.5 is the recorded systolic/diastolic pressure.
- If the two pressure measurements <u>differ by more than 5 mmHg</u>, then a third reading measurement is made, and the average of the three becomes the recorded pressure. For example, if the three measurements are 115/90, 124/96, and 120/92, then 119.7/92.7 is the recorded systolic/diastolic pressure. The recorded blood pressure will be the average of the measurements.
- Record the heart rate. For heart rate, the average of the two (or three, if performed) measurements obtained becomes the recorded heart rate.

#### 21.4.4. EKG

EKGs will be recorded at Screening (Day -7 to Day -1) and reviewed for abnormalities by the Clinical Investigator prior to enrollment. EKGs will also be performed at Visit 3 (Day  $8 \pm 1$ ), Visit 5 (Day  $30\pm 2$ ), and Visit 8/Exit (Day  $90\pm 3$ ).

# 21.4.5. Best Corrected Visual Acuity

ETDRS chart will be used to examine BCVA at each study visit. See Study Procedures manual for the detailed procedure for measuring visual acuity.

# 21.4.6. Slit-Lamp Biomicroscopy

Slit-lamp biomicroscopy will be used to examine eye structures at each study visit. Slit-lamp biomicroscopy will be performed prior to injection and then again within 30 minutes after injection on the visit of DE-122 or anti-VEGF injection.

The lid, conjunctiva, cornea, and lens will be observed with the slit-lamp beam approximately 0.3 mm in width and 1.0 mm in length and graded on a 4-point scale (0-3 scale) as described below:

## **Lid Redness**

None (0) = Normal

Mild (1) = Redness of most or all the lid(s) margin OR skin

Moderate (2) = Redness of most or all the lid(s) margin AND skin

Severe (3) = Marked diffuse redness of both lid(s) margin AND skin

### Lid Edema

None (0) = Normal

Mild (1) = Localized to a small region of the lid(s)

Moderate (2) = Diffuse, most or all the lid(s) but not prominent/protruding

Severe (3) = Diffuse, most or all the lid(s) AND prominent/protruding

# Conjunctival (Palpebral and Bulbar) Hyperemia

None (0) = Normal

Mild (1) = Slight localized injection

Moderate (2) = Pink color, confined to palpebral OR bulbar conjunctiva

Severe (3) = Red color of the palpebral AND/OR bulbar conjunctiva

# **Conjunctival Edema**

None (0) = Normal

Mild (1) = Slight localized swelling

Moderate (2) = Mild/medium localized swelling or mild diffuse swelling

Severe (3) = Moderate diffuse swelling

## **Corneal Edema**

None (0) = Normal

Mild (1) = Mild, diffuse stromal haze

Moderate (2) = Dense, diffuse stromal haze or bullae

Severe (3) = Dense, diffuse bullae or stromal haze AND stromal edema

#### Lens

The lens will be noted as phakic, aphakic, or pseudophakic. Phakic lens will be graded as described below:

None (0) = No lens discoloration nor opacification

Mild (1) = Yellow lens discoloration or small lens opacity (axial or peripheral)

Moderate (2) = Amber lens discoloration or medium lens opacity (axial or peripheral)

Severe (3) = Brunescent lens discoloration or complete lens opacification (no red reflex)

Anterior chamber cells and flare will be observed with a 1.0 mm in width and 1.0 mm in length slit beam and graded using the Standardization of Uveitis Nomenclature (SUN) scale (Sun Working Group, 2005). The iris and the pupil will be evaluated for the presence of clinically significant abnormalities.

## **Anterior Chamber Cells**

- (0) = No cells
- (0.5) = 1-5 cells
- (1) = 6-15 cells
- (2) = 16-25 cells
- (3) = 26-50 cells

(4) = >50 cells

### **Anterior Chamber Flare**

- (0) = None
- (1) = Faint
- (2) = Moderate (iris/lens details clear)
- (3) = Marked (iris/lens details hazy)
- (4) = Intense (fibrin/plastic aqueous)

#### **Iris**

The iris will be evaluated for the presence of any clinically significant abnormalities, and graded as either normal (within normal limits) or abnormal (clinically significant abnormality present). A description of any clinically significant abnormalities will be noted.

# Pupil

The pupil will be evaluated for the presence of any clinically significant abnormalities, and graded as either normal (within normal limits) or abnormal (clinically significant abnormality present). A description of any clinically significant abnormalities will be noted.

#### 21.4.7. Intraocular Pressure

IOP will be measured by applanation tonometry at each study visit. At the visit of DE-122 or anti-VEGF medication injection, IOP will be measured before DE-122 or anti-VEGF medication injection and 40 ( $\pm 10$ ) minutes after injection. If post-injection IOP is increased  $\geq 10$  mmHg from pre-injection IOP, the IOP will be measured again 60 ( $\pm 10$ ) minutes following injection. If there is an increase of  $\geq 10$  mmHg at 60 ( $\pm 10$ ) minutes post-injection compared to pre-injection IOP, the subject will be prescribed a topical IOP-lowering medication until he or she returns for follow-up per the Clinical Investigator's discretion (an unscheduled visit may apply), and the IOP increase of  $\geq 10$  mmHg shall be reported as an AE.

## IOP should be measured only after the biomicroscopy examination has been completed.

The applanation tonometer must be calibrated for accuracy before the first subject undergoes screening, and periodically until the last subject has exited the study. For checking calibration, follow the manufacturer's instructions.

The following IOP measurement procedure is in accordance with the procedure used in the Ocular Hypertension Treatment Study (Gordon et al., 2001) at each visit:

The right eye is always tested first. At least two, and sometimes three, consecutive measurements are made to obtain a determination of intraocular pressure. Each IOP measurement should be recorded in the subject's source document and in the eCRFs.

• If the two measurements differ by 2 mmHg or less, then the average of the two measurements becomes the recorded IOP. For example, if the two measurements are 22 and 23, then 22.5 is the final recorded IOP.

- However, if the two measurements differ by 3 mmHg or more, then a third measurement is made, and the median of the three measurements becomes the recorded IOP (the median is the middle measurement after arraying the measurements from low to high). For example, if the three measurements are 15, 19, and 16, then 16 is the final recorded IOP.
- The IOP in the left eye is then measured using the same technique.

# 21.4.8. Indirect Ophthalmoscopy

Indirect ophthalmoscopy will be performed for each eye at each visit with pupil dilation.

Indirect ophthalmoscopy will be used to examine the retina at each study visit. Indirect ophthalmoscopy will be performed prior to and within 30 minutes after each DE-122 or anti-VEGF medication injection. Areas to be assessed include cup to disc ratio, retina, macula and choroid, and vitreous.

## Cup/Disc Ratio

The cup/disc ratio will be determined by the examiner and recorded using two decimal places (e.g., 0.80).

# Retina, Macula and Choroid

The retina, macula and choroid will be evaluated for the presence of any clinically significant abnormalities, and graded as either normal (within normal limits) or abnormal (clinically significant abnormality present). A description of any abnormalities will be noted.

#### Vitreous

The following National Eye Institute Grading Scheme will be used to measure vitreous haze and opacification (Nussenblatt et al., 1985).

#### Vitreous Haze Scale

| Step | Description |
|-----------------|---------------------------------------------|
| (0) | Clear |
| (Trace or 0.5+) | Trace |
| (1+) | Few opacities, mild blurring |
| (2+) | Significant blurring but still visible |
| (3+) | Optic nerve visible, no vessels seen |
| (4+) | Dense opacity obscures the optic nerve head |

# 21.4.9. Spectral Domain Optical Coherence Tomography

Spectralis, Cirrus or 3D OCT will be utilized to take optical images of both eyes at each study visit. The same machine must be used consistently throughout the study for any given subject.

### 21.4.10. Fundus Photography

Digital color fundus photography will be taken at Screening (Day -7 to Day -1), Visit 5 (Day 30±2), Visit 7 (Day 60±3) and Visit 8/Exit (Day 90±3) in both eyes. Required fields to be captured are:

- The optic disc, Field 1
- The macula, Field 2

# 21.4.11. Fluorescein Angiography

Fundus fluorescein angiography will be taken at Screening (Day -7 to Day -1), Visit 5 (Day 30±2), Visit 7 (Day 60±3) and Visit 8/Exit (Day 90±3) in both eyes. Required fields to be captured are:

- The optic disc, Field 1
- The macula, Field 2

# 21.4.12. Urine Pregnancy Test

A urine pregnancy test will be conducted at Visit 5 (Day 30±2) and Visit 7 (Day 60±3) for all women of childbearing potential. A female is considered of childbearing potential unless she is post-menopausal (at least 24 months since last menses occurred), has had her uterus and/or both ovaries removed, or has had a bilateral tubal ligation. To obtain the pregnancy test, the subject should follow instructions provided by the manufacturer of the urine pregnancy test kit.

# 21.4.13. Serum Pregnancy Test

A serum pregnancy test will be conducted at Screening (Day -7 to Day -1) and Visit 8/Exit (Day 90±3) for all women of childbearing potential. A female is considered of childbearing potential unless she is post-menopausal (at least 24 months since last menses occurred), has had her uterus and/or both ovaries removed, or has had a bilateral tubal ligation. To perform the pregnancy test, Human chorionic gonadotropin (hCG) will be contained into serum parameters that will be measured.

## 21.4.14. Hematology, Chemistry and Urinalysis

Approximately 10 mL of fasting blood and urine samples will be obtained at Screening (Day -7 to Day -1), Visit 3(Day 8±1), Visit 5 (Day 30±2) and Visit 8/Exit (Day 90±3). The subjects will be asked to fast for a minimum of 8 hours prior to each blood and urine collection. Samples will be sent to a central laboratory for analysis.

# Serum Chemistry, Hematology

The following is a list of the minimum parameters that will be measured. Other additional parameters may also be reported.

| Chemistry | Hematology |
|---|---|
| Albumin | red blood cells (RBC) |
| Creatinine | white blood cells (WBC) |
| lactate dehydrogenase (LDH) | differential WBC |
| glucose | platelets (PLT) |
| calcium | hemoglobin (HGB) |
| potassium | hematocrit (HCT) |
| sodium | mean corpuscular volume (MCV) |
| cholesterol (total, HDL and LDL) | mean corpuscular hemoglobin (MCH) |
| triglycerides | mean corpuscular hemoglobin conc. (MCHC) |
| urea nitrogen | |
| bilirubin (total, direct, indirect) | |
| alkaline phosphatase (ALP) | |
| alanine aminotransferase (ALT) | |
| aspartate aminotransferase (AST) | |
| gamma glutamyl transferase (GGT) | |
| Human chorionic gonadotropin (hCG)* | |

Prior to enrolling a subject, the Clinical Investigator will indicate on the source document if any screening laboratory values exclude the subject from participating in the study (e.g., serum creatinine > 1.3 mg/dL).

# Urinalysis

The following is a list of the minimum urine parameters that will be measured. Other additional urine parameters may also be reported.

| Urinalysis |
|--------------|
| PH |
| Protein |
| Erythrocytes |
| Ketones |
| Glucose |

<sup>\*</sup>conduct only at Screening (Day -7 to Day -1) and Visit 8/Exit (Day 90±3).

Prior to enrolling a subject, the Clinical Investigator will indicate on the source document if any screening laboratory values exclude the subject from participating in the study.

# 21.4.15. Procedure for Immunogenicity Serum Sample

Approximately 5 mL of serum sample will be collected for immunogenicity analysis from the subject at Visit 1 (Day 1) and Visit 5 (Day 30±2).

Refer to the separate procedure manual for sample handling, storage, and shipment.

# 21.4.16. Procedure for Biomarker Serum Sample

Approximately 10 mL of blood sample will be collected for biomarker analysis from the subject at Visit 1 (Day 1), Visit 2 (Day 2), Visit 3 (Day 8±1), Visit 5 (Day 30±2) and Visit 8 (Day 90±3).

There will be up to 5 blood draws for Biomarker. The total amount of blood collected from each subject in Cohort 3 and Cohort 4 during this study will be approximately 50 mL.

Refer to the separate procedure manual for sample handling, storage, and shipment.

 Table 6:
 Protocol Amendment 03 Summary of Changes

| Page | Section Number and Title | Description of Change |
|---|---|---|
| 4-8 | 2.SYNOPSIS | Modifications were made to reflect the study period and the study design changes made throughout the protocol. |
| 16 | 5. INTRODUCTION | Rationale: To update the status of the study. Amendment 02 text: (None) Amendment 03 text: As of June 2016, 2 subjects in Cohort 1 have been |
| | | enrolled and completed the study with no adverse events, and no safety and tolerability concerns. |
| 19 | 7.1. Overall Study Design and Plan. | Rationale: To allow the cohort transition from Cohort 1 to Cohort 2 with 2 subjects safety data at least, according to the upadated study status. Amendment 02 context: Three subjects will be enrolled in Cohort 1. Three subjects safety data is required to make a decision by Safety Review Team whether or not the transition to Cohort 2 is acceptable. Amendment 03 context: Two or Three subjects will be enrolled in Cohort 1. Two subjects safety data at least is required to make a decision by Safety Review Team whether or not the transition to Cohort 2 is acceptable. |
| 20 | Figure 1: Study Shematic | Rationale: Updated in accordance with the change of overall study design and plan. |
| 21 | 7.2. Number of Subjects | Rationale: In accordance with the change of overall study design and plan and change of number of sites. Amendment 02 text: Approximately 12 subjects (3 subjects per cohort) with refractory exudative age related macular degeneration will be enrolled at 3-4 sites. Amendment 03 text: Approximately 12 subjects (2 or 3 subjects in Cohort 1, 3 subjects each in Cohorts 2, 3 and 4) with refractory exudative age related macular degeneration will be enrolled at 5 sites. |
| 22 | 7.4. Dose Adjustment Criteria | Rationale: In accordance with the change of overall study design. Amendment 02 text: When all subjects in the cohort have completed Visit 5 (Day 30±2), the Safety Review Team will again evaluate the safety parameters. Amendment 03 text: When the first 2 or 3 subjects in Cohort 1 and 3 subjects in other Cohorts have completed Visit 5 (Day 30±2), the Safety Review Team will again evaluate the safety parameters. |

**Table 6:** Protocol Amendment 03 Summary of Changes (Continued)

| Page | Section Number and Title | Description of Change |
|---|---|---|
| 24 | Table 4: Schedule of Events | Rationale: Updated in accordance with the addition of blood sample collection for biomarker analysisis. |
| 25 | 7.6.2.1. Visit 1 (Day 1) | Rationale: To add blood sample collection for |
| 27 | 7.6.2.2. Visit 2 (Day 2) | biomarker analysis. |
| 27 | 7.6.2.3. Visit 3 (Day 8±1) | Amendment 02 text: |
| 29 | 7.6.2.5. Visit 5 (Day 30±2) | (None) |
| 31 | 7.6.3.1. Visit 8/Exit (Day | Amendment 03 text: |
| | 90±3) | Biomarker serum sample (in Cohorts 3 and 4) |
| 33 | 8.1. Subjects Inclusion Criteria | Rationale: To expand the subjects enrollment according to the updated status of the study in which no safety issue was seen so far. Amendment 02 text: |
| | | 8.BCVA of 50 to 20 ETDRS letters (20/100 to |
| | | 20/400) in the study eye. |
| | | Amendment 03 text: |
| | | 8.BCVA of 65 to 20 ETDRS letters (20/50 to |
| | | 20/400) in the study eye. |
| 51 | 13. OTHER ASSESSMENTS | Rationale: To add biomarker analysis. |
| | | Amendment 02 text: |
| | | 13.3 Other Assessments |
| | | Other assessments include concomitant |
| | | medications and exposure to study drug. |
| | | Amendment 03 text: 13.3 Biomarker |
| | | For the biomarker finding, serum samples will be collected according examination schedule from the |
| | | subjects in Cohorts 3 and 4, and measured for |
| | | levels of endoglin-related proteins. The remaining |
| | | serum samples will be stored for future exploratory |
| | | research to identify possible other biomarkers |
| | | associated with the study drug(s) and/or |
| | | ophthalmologic disease conditions. |
| | | 13.4 Other Assessments |
| | | Other assessments include concomitant |
| | | medications and exposure to study drug. |

**Table 6:** Protocol Amendment 03 Summary of Changes (Continued)

| Page | Section Number and Title | Description of Change |
|---|---|---|
| 52 | 14.1.2. Sample Size | Rationale: In accordance with the change of overall study design and plan and change of number or sites. Amendment 02 text: Approximately 12 subjects (3 subjects per cohort) with refractory exudative age related macular degeneration will be enrolled at 3-4 sites. Amendment 03 text: Approximately twelve subjects (2 or 3 subjects in Cohort 1; 3 subjects in Cohorts 2, 3, and 4) with refractory exudative age related macular degeneration will be enrolled at 5 sites. |
| 54 | 14.8.2. Biomarker Analysis | Rationale: To add biomarker analysis. Amendment 02 text: (None) Amendment 03 text: Changes from baseline in levels of biomarkers will be summarized descriptively by dose level of DE-122. |
| 81 | 24.1.16. Procedure for Biomarker Serum Sample | Rationale: To add biomarker analysis. Amendment 02 text: (None) Amendment 03 text: Approximately 10 mL of blood sample will be collected for biomarker analysis from the subject at Visit 1 (Day 1), Visit 2 (Day 2), Visit 3 (Day 8±1), Visit 5 (Day 30±2) and Visit 8 (Day 90±3). There will be up to approximately 5 blood draws for Biomarker. The total amount of blood collected from each subject in Cohort 3 and Cohort 4 during this study will be up to approximately 50 mL. Refer to the separate procedure manual for sample handling, storage, and shipment. |